CLINICAL TRIAL: NCT01381575
Title: Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' HPV-16/18 L1 AS04 Vaccine When Administered According to Alternative 2-dose Schedules in 9 - 14 Year Old Females
Brief Title: Evaluation of Immunogenicity and Safety of Two 2-dose Human Papillomavirus (HPV) Vaccine Schedules in 9-14 Year Old Girls
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114700; 2011-000757-22 (EudraCT Number)
Record Dates: First submitted 2011-06-17; First posted 2011-06-27 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Infections, Papillomavirus
Keywords: HPV infection; Human Papillomavirus; Cervical cancer; HPV-16; HPV-18; vaccine
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18

ARMS (3):
- Cervarix 1 Group (Experimental): Female subjects aged 9 to 14 years at the time of the first vaccination, who received 2 doses of the Cervarix vaccine at Day 0 and at Month 6, respectively. The vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm.
  Interventions: Biological: GSK Biologicals' HPV vaccine 580299
- Cervarix 2 Group (Active Comparator): Female subjects aged 15 to 25 years at the time of the first vaccination, who received 3 doses of the Cervarix vaccine at Day 0, at Month 1 and at Month 6, respectively. The vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm.
  Interventions: Biological: GSK Biologicals' HPV vaccine 580299
- Cervarix 3 Group (Experimental): Female subjects aged 9 to 14 years at the time of the first vaccination, who received 2 doses of the Cervarix vaccine at Day 0 and at Month 12, respectively. The vaccine was administered intramuscularly into the deltoid muscle of the non-dominant arm.
  Interventions: Biological: GSK Biologicals' HPV vaccine 580299

INTERVENTIONS:
Biological: GSK Biologicals' HPV vaccine 580299 — Subjects received 2 or 3 doses of HPV vaccine administered intramuscularly.
  Other Names: Cervarix

SUMMARY:
This study has been designed to evaluate the immunogenicity and safety of GSK Biologicals' HPV-16/18 vaccine when administered according to alternative 2-dose schedules (0,6 months and 0,12 months) in healthy 9-14 year old females as compared to the standard 3-dose schedule (0,1,6 months) in 15-25 year old females.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol or/ and subjects who the investigator believes their parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol
* A female between, and including, 9 and 25 years of age at the time of the first vaccination
* Written informed consent obtained from the subject/from the parent(s)/LAR(s) of the subject prior to enrolment in the study. In addition, subjects below the legal age of consent should sign and personally date a written informed assent form
* Healthy subjects
* Female subjects of non-childbearing potential may be enrolled in the study
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire vaccination period and up to two months after the last study vaccine dose

Exclusion Criteria:

* Pregnant or breastfeeding
* A female planning to become pregnant, likely to become pregnant or planning to discontinue contraceptive precautions during the entire vaccination period and up to two months after the last study vaccine dose
* Previous vaccination against HPV or planned administration of another HPV vaccine during the study
* Child in care. A child in care is a child who has been placed under the control or protection of an agency, organisation, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. The definition of a child in care does not include a child who is adopted or has an appointed legal guardian.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccines
* Cancer or autoimmune disease under treatment
* Planned administration/administration of a vaccine/product not foreseen by the study protocol within 30 days before each dose of vaccine. Administration of routine meningococcal, hepatitis B, hepatitis A, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus-containing vaccine up to 8 days before each dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Previous administration of MPL or AS04 adjuvant.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition
* Family history of congenital or hereditary immunodeficiency
* Major congenital defects or serious chronic illness
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests, which in the opinion of the investigator precludes administration of the study vaccine
* Acute disease and/or fever at the time of enrolment

Ages: 9 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1447 (Actual)
Dates: Start 2011-06-29 (Actual); Primary Completion 2012-06-28 (Actual); Study Completion 2014-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- Canada (6):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Woodstock, Ontario
  - GSK Investigational Site, Sherbrooke, Quebec
- Germany (14):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Schönau am Königssee, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Wolfsburg, Lower Saxony
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Weimar, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (6):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Cuneo, Piedmont
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Ragusa, Sicily
  - GSK Investigational Site, Padua, Veneto
- Taiwan (2):
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=4511

REFERENCES:
- [Background] Huang LM, Puthanakit T, Cheng-Hsun C, Ren-Bin T, Schwarz T, Pellegrino A, Esposito S, Frenette L, McNeil S, Durando P, Rheault P, Giaquinto C, Horn M, Petry KU, Peters K, Azhar T, Hillemanns P, De Simoni S, Friel D, Pemmaraju S, Hezareh M, Thomas F, Descamps D, Folschweiller N, Struyf F. Sustained Immunogenicity of 2-dose Human Papillomavirus 16/18 AS04-adjuvanted Vaccine Schedules in Girls Aged 9-14 Years: A Randomized Trial. J Infect Dis. 2017 Jun 1;215(11):1711-1719. doi: 10.1093/infdis/jix154. PMID 28591778
- [Background] Puthanakit T, Huang LM, Chiu CH, Tang RB, Schwarz TF, Esposito S, Frenette L, Giaquinto C, McNeil S, Rheault P, Durando P, Horn M, Klar M, Poncelet S, De Simoni S, Friel D, De Muynck B, Suryakiran PV, Hezareh M, Descamps D, Thomas F, Struyf F. Randomized Open Trial Comparing 2-Dose Regimens of the Human Papillomavirus 16/18 AS04-Adjuvanted Vaccine in Girls Aged 9-14 Years Versus a 3-Dose Regimen in Women Aged 15-25 Years. J Infect Dis. 2016 Aug 15;214(4):525-36. doi: 10.1093/infdis/jiw036. Epub 2016 Feb 3. PMID 26908726
- [Background] Stevenson L, Huang LM, Berlaimont V, Folschweiller N. Reply to Poddighe. J Infect Dis. 2017 Sep 15;216(6):783-785. doi: 10.1093/infdis/jix365. No abstract available. PMID 28934440
- [Background] Folschweiller N, Behre U, Dionne M, Durando P, Esposito S, Ferguson L, Ferguson M, Hillemanns P, McNeil SA, Peters K, Ramjattan B, Schwarz TF, Supparatpinyo K, Suryakirian PV, Janssens M, Moris P, Decreux A, Poncelet S, Struyf F. Long-term Cross-reactivity Against Nonvaccine Human Papillomavirus Types 31 and 45 After 2- or 3-Dose Schedules of the AS04-Adjuvanted Human HPV-16/18 Vaccine. J Infect Dis. 2019 May 5;219(11):1799-1803. doi: 10.1093/infdis/jiy743. PMID 30715452
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 114700 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114700 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114700 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114700 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114700 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114700 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by 33 principal investigators in five countries (Canada, Germany, Italy, Taiwan and Thailand).
Pre-assignment Details: All 1447 subjects enrolled in the study were vaccinated and included in the Total vaccinated cohort (TVC).
Period: Overall Study
Arm/Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group
Started | 550 | 482 | 415
Completed | 524 | 443 | 395
Not Completed | 26 | 39 | 20
Not completed — Serious Adverse Event | 1 | 0 | 0
Not completed — Non-Serious Adverse Event | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 15 | 9 | 7
Not completed — Migrated/moved from study area | 2 | 12 | 2
Not completed — Lost to Follow-up | 8 | 17 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Total
Number analyzed (Participants) | 550 | 482 | 415 | 1447
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.6 (1.59) | 19.6 (3.05) | 11.4 (1.55) | 14.2 (4.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 550 | 482 | 415 | 1447
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 6 | 3 | 6 | 15
  Asian - Central/South Asian Heritage | 1 | 1 | 4 | 6
  Asian - East Asian Heritage | 141 | 105 | 74 | 320
  Asian - South East Asian Heritage | 108 | 106 | 104 | 318
  White - Arabic / North African Heritage | 1 | 0 | 1 | 2
  White - Caucasian / European Heritage | 288 | 263 | 223 | 774
  Mixed origin | 5 | 4 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies in Cervarix 1 Group and Cervarix 2 Group at Month 7
Description: Seroconversion was defined as the appearance of antibodies (anti-HPV-16 concentrations greater than or equal to (≥) 8 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL) and anti-HPV-18 concentrations ≥ 7 EL.U/mL) in the serum of subjects seronegative before vaccination. A seronegative subject was a subject with anti-HPV-16/18 antibody concentration lower than (<) 8/7 EL.U/mL, respectively.
Time Frame: At Month 7 (i.e. one month after the last dose of study vaccine)
Population: The analysis was based on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available, who were seronegative before vaccination and for whom assay results were available for antibodies against at least one study vaccine antigen component at Month 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1 Group | Cervarix 2 Group
Number analyzed (Participants) | 493 | 382
Participants
  Anti-HPV-16: number analyzed (Participants) | 488 | 352
  Anti-HPV-16 | 488 | 352
  Anti-HPV-18 | 493 | 382
Statistical Analysis 1: Comparison: Cervarix 1 Group vs Cervarix 2 Group; Immune response to anti-HPV-16 in terms of seroconversion (SCR) rates: To evaluate sequentially if the immunogenicity (as determined by ELISA) of Cervarix vaccine administered according to a 2-dose schedule of 0,6 months in 9-14 year old females was non-inferior to that administered according to the standard 3-dose schedule of 0,1,6 months in 15-25 year old females, 1 month after the last dose of study vaccine, in initially seronegative subjects; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion was demonstrated if, 1 month after the last dose, for both anti-HPV-16 and anti-HPV-18, the upper limit of the 95% Confidence Interval (CI) for the difference (Cervarix 2 Group minus Cervarix 1 Group) was below 5%; Difference in SCR = 0.0, 95% CI 2-sided [-1.08 to 0.78]
Statistical Analysis 2: Comparison: Cervarix 1 Group vs Cervarix 2 Group; Immune response to anti-HPV-18 in terms of seroconversion (SCR) rates: To evaluate sequentially if the immunogenicity (as determined by ELISA) of Cervarix vaccine administered according to a 2-dose schedule of 0,6 months in 9-14 year old females was non-inferior to that administered according to the standard 3-dose schedule of 0,1,6 months in 15-25 year old females, 1 month after the last dose of study vaccine, in initially seronegative subjects; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in SCR = 0.0, 95% CI 2-sided [-1.00 to 0.77]

2. Primary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Concentrations (by ELISA) in Cervarix 1 Group and Cervarix 2 Group at Month 7
Description: Antibody concentrations were assessed by ELISA and expressed as geometric mean concentrations (GMCs) in EL.U/mL.
Time Frame: At Month 7 (i.e. one month after the last dose of study vaccine)
Population: The analysis was based on the ATP cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available, who were seronegative before vaccination and for whom assay results were available for antibodies against at least one study vaccine antigen component at Month 7.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 1 Group | Cervarix 2 Group
Number analyzed (Participants) | 493 | 382
EL.U/mL
  Anti-HPV-16: number analyzed (Participants) | 488 | 352
  Anti-HPV-16 | 9400.1 [8818.3 to 10020.4] | 10234.5 [9258.3 to 11313.6]
  Anti-HPV-18 | 5909.1 [5508.9 to 6338.4] | 5002.6 [4572.6 to 5473.1]
Statistical Analysis 1: Comparison: Cervarix 1 Group vs Cervarix 2 Group; Immune response to anti-HPV-16 in terms of Geometric Mean Concentrations (GMCs): To evaluate sequentially if the immunogenicity (as determined by ELISA) of Cervarix vaccine administered according to a 2-dose schedule at 0, 6 months in 9-14 year old females was non-inferior to that administered according to the standard 3-dose schedule of 0,1,6 months in 15-25 year old females, 1 month after the last dose of study vaccine, in initially seronegative subjects; Test type: Non-Inferiority — Non-inferiority with respect to Geometric Mean Concentrations (GMCs) was demonstrated if, 1 month after the last dose, for both anti-HPV-16 and anti-HPV-18, the upper limit of 95% CI for the GMT ratio (Cervarix 2 Group divided by Cervarix 1 Group) was below 2; Geometric mean ratio = 1.09, 95% CI 2-sided [0.97 to 1.22]
Statistical Analysis 2: Comparison: Cervarix 1 Group vs Cervarix 2 Group; Immune response to anti-HPV-18 in terms of Geometric Mean Concentrations (GMCs): To evaluate sequentially if the immunogenicity (as determined by ELISA) of Cervarix vaccine administered according to a 2-dose schedule at 0, 6 months in 9-14 year old females was non-inferior to that administered according to the standard 3-dose schedule of 0,1,6 months in 15-25 year old females, 1 month after the last dose of study vaccine, in initially seronegative subjects; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 0.85, 95% CI 2-sided [0.76 to 0.95]

3. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-16 and Anti-HPV-18 Antibodies in Cervarix 1 Group and Cervarix 2 Group at Day 0 and at Months 7, 12, 18, 24 and 36
Description: Seroconversion was defined as the appearance of antibodies (anti-HPV-16 concentrations ≥ 8 EL.U/mL and anti-HPV-18 concentrations ≥ 7 EL.U/mL [applicable for Day 0, Month 7 and Month 12 time points] and anti-HPV-16 concentrations ≥ 19 EL.U/mL and anti-HPV-18 concentrations ≥ 18 EL.U/mL [applicable for Month 18, Month 24 and Month 36 time points]) in the serum of subjects seronegative before vaccination.
  A seronegative subject was a subject with an anti-HPV-16/18 antibody concentration below (<) the aforementioned cut-offs.
  Note: In order to increase the ELISA precision, the assay cut-off value was changed from 8 EL.U/mL to 19 EL.U/mL for HPV-16 and from 7 EL.U/mL to 18 EL.U/mL for HPV-18 from Month 18 onwards.
Time Frame: At Day 0 and at Months 7, 12, 18, 24 and 36
Population: The analysis was based on the Month 36 ATP cohort for immunogenicity which included all subjects seronegative before vaccination, who returned for blood sampling at Month 36 and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination at the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1 Group | Cervarix 2 Group
Number analyzed (Participants) | 462 | 356
Participants
  Anti-HPV-16, Day 0: number analyzed (Participants) | 455 | 330
  Anti-HPV-16, Day 0 | 0 | 0
  Anti-HPV-16, Month 7: number analyzed (Participants) | 455 | 330
  Anti-HPV-16, Month 7 | 455 | 330
  Anti-HPV-16, Month 12: number analyzed (Participants) | 455 | 330
  Anti-HPV-16, Month 12 | 455 | 330
  Anti-HPV-16, Month 18: number analyzed (Participants) | 453 | 329
  Anti-HPV-16, Month 18 | 453 | 329
  Anti-HPV-16, Month 24: number analyzed (Participants) | 454 | 326
  Anti-HPV-16, Month 24 | 454 | 326
  Anti-HPV-16, Month 36: number analyzed (Participants) | 455 | 330
  Anti-HPV-16, Month 36 | 455 | 330
  Anti-HPV-18, Day 0 | 0 | 0
  Anti-HPV-18, Month 7 | 462 | 356
  Anti-HPV-18, Month 12 | 462 | 356
  Anti-HPV-18, Month 18: number analyzed (Participants) | 459 | 355
  Anti-HPV-18, Month 18 | 458 | 355
  Anti-HPV-18, Month 24: number analyzed (Participants) | 460 | 352
  Anti-HPV-18, Month 24 | 459 | 352
  Anti-HPV-18, Month 36 | 461 | 355

4. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Concentrations (by ELISA) in Cervarix 1 Group and Cervarix 2 Group at Day 0 and at Months 7, 12, 18, 24 and 36
Description: Antibody concentrations were assessed by ELISA and expressed as geometric mean concentrations (GMCs) in EL.U/mL.
Time Frame: At Day 0 and at Months 7, 12, 18, 24 and 36
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 1 Group | Cervarix 2 Group
Number analyzed (Participants) | 462 | 356
EL.U/mL
  Anti-HPV-16, Day 0: number analyzed (Participants) | 455 | 330
  Anti-HPV-16, Day 0 | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  Anti-HPV-16, Month 7: number analyzed (Participants) | 455 | 330
  Anti-HPV-16, Month 7 | 9402.9 [8792.4 to 10055.8] | 10120.2 [9162.7 to 11177.9]
  Anti-HPV-16, Month 12: number analyzed (Participants) | 455 | 330
  Anti-HPV-16, Month 12 | 2653.5 [2473.5 to 2846.6] | 3290.4 [2956.5 to 3662.0]
  Anti-HPV-16, Month 18: number analyzed (Participants) | 453 | 329
  Anti-HPV-16, Month 18 | 1730.7 [1608.6 to 1862.0] | 1931.2 [1735.4 to 2149.1]
  Anti-HPV-16, Month 24: number analyzed (Participants) | 454 | 326
  Anti-HPV-16, Month 24 | 1483.8 [1382.1 to 1592.9] | 1575.9 [1418.2 to 1751.2]
  Anti-HPV-16, Month 36: number analyzed (Participants) | 455 | 330
  Anti-HPV-16, Month 36 | 1210.2 [1124.8 to 1302.1] | 1326.4 [1193.9 to 1473.5]
  Anti-HPV-18, Day 0 | 3.5 [3.5 to 3.5] | 3.5 [3.5 to 3.5]
  Anti-HPV-18, Month 7 | 5935.6 [5519.4 to 6383.3] | 4984.2 [4543.9 to 5467.1]
  Anti-HPV-18, Month 12 | 1523.6 [1403.7 to 1653.7] | 1491.5 [1339.0 to 1661.4]
  Anti-HPV-18, Month 18: number analyzed (Participants) | 459 | 355
  Anti-HPV-18, Month 18 | 864.6 [793.1 to 942.7] | 830.6 [742.9 to 928.5]
  Anti-HPV-18, Month 24: number analyzed (Participants) | 460 | 352
  Anti-HPV-18, Month 24 | 715.5 [658.1 to 777.9] | 654.3 [582.9 to 734.5]
  Anti-HPV-18, Month 36 | 562.8 [516.4 to 613.4] | 552.6 [494.1 to 618.0]

5. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-16 and Anti-HPV-18 Antibodies in Cervarix 3 Group
Description: Seroconversion was defined as the appearance of antibodies (anti-HPV-16 concentrations ≥ 8 EL.U/mL and anti-HPV-18 concentrations ≥ 7 EL.U/mL [applicable for Day 0 and Month 13 time points] and anti-HPV-16 concentrations ≥ 19 EL.U/mL and anti-HPV-18 concentrations ≥ 18 EL.U/mL [applicable for Month 18, Month 24 and Month 36 time points]) in the serum of subjects seronegative before vaccination.
  A seronegative subject was a subject with an anti-HPV-16/18 antibody concentration below (<) the aforementioned cut-offs.
  Note: In order to increase the ELISA precision, the assay cut-off value was changed from 8 EL.U/mL to 19 EL.U/mL for HPV-16 and from 7 EL.U/mL to 18 EL.U/mL for HPV-18 from Month 18 onwards.
Time Frame: At Day 0 and at Months 13, 18, 24 and 36
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 3 Group
Number analyzed (Participants) | 355
Participants
  Anti-HPV-16, Day 0: number analyzed (Participants) | 339
  Anti-HPV-16, Day 0 | 0
  Anti-HPV-16, Month 13: number analyzed (Participants) | 339
  Anti-HPV-16, Month 13 | 339
  Anti-HPV-16, Month 18: number analyzed (Participants) | 339
  Anti-HPV-16, Month 18 | 339
  Anti-HPV-16, Month 24: number analyzed (Participants) | 337
  Anti-HPV-16, Month 24 | 337
  Anti-HPV-16, Month 36: number analyzed (Participants) | 339
  Anti-HPV-16, Month 36 | 339
  Anti-HPV-18, Day 0 | 0
  Anti-HPV-18, Month 13 | 355
  Anti-HPV-18, Month 18 | 355
  Anti-HPV-18, Month 24: number analyzed (Participants) | 353
  Anti-HPV-18, Month 24 | 353
  Anti-HPV-18, Month 36 | 355

6. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Concentrations (by ELISA) in Cervarix 3 Group
Description: Antibody concentrations were assessed by ELISA and expressed as geometric mean concentrations (GMCs) in EL.U/mL.
Time Frame: At Day 0 and at Months 13, 18, 24 and 36
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix 3 Group
Number analyzed (Participants) | 355
EL.U/mL
  Anti-HPV-16, Day 0: number analyzed (Participants) | 339
  Anti-HPV-16, Day 0 | 4.0 [4.0 to 4.0]
  Anti-HPV-16, Month 13: number analyzed (Participants) | 339
  Anti-HPV-16, Month 13 | 11329.4 [10509.3 to 12213.5]
  Anti-HPV-16, Month 18: number analyzed (Participants) | 339
  Anti-HPV-16, Month 18 | 3248.2 [2974.2 to 3547.4]
  Anti-HPV-16, Month 24: number analyzed (Participants) | 337
  Anti-HPV-16, Month 24 | 2191.0 [2003.9 to 2395.5]
  Anti-HPV-16, Month 36: number analyzed (Participants) | 339
  Anti-HPV-16, Month 36 | 1559.3 [1431.2 to 1699.0]
  Anti-HPV-18, Day 0 | 3.5 [3.5 to 3.5]
  Anti-HPV-18, Month 13 | 6580.0 [6075.8 to 7126.0]
  Anti-HPV-18, Month 18 | 1860.3 [1699.4 to 2036.4]
  Anti-HPV-18, Month 24: number analyzed (Participants) | 353
  Anti-HPV-18, Month 24 | 1174.7 [1067.1 to 1293.2]
  Anti-HPV-18, Month 36 | 804.0 [731.8 to 883.4]

7. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Titers [by Pseudovirion-Based Neutralisation Assay (PBNA)] in a Subset of Subjects From Cervarix 3 Group
Description: Antibody titers were expressed as geometric mean titers (GMTs). The cut-off of the assay was 40 ED50 for both anti-HPV-16 and anti-HPV-18. The assay was performed on a subset of 100 subjects from Cervarix 3 Group.
Time Frame: At Day 0 and at Months 13, 18, 24 and 36
Population: The analysis was based on the Month 36 ATP cohort for immunogenicity which included a subset of 100 subjects from Cervarix 3 Group, who returned for blood sampling at Month 36 and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination at the specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix 3 Group
Number analyzed (Participants) | 88
Titers
  Anti-HPV-16, Day 0 | 20.0 [20.0 to 20.0]
  Anti-HPV-16, Month 13 | 74848.0 [60521.9 to 92565.1]
  Anti-HPV-16, Month 18 | 16576.6 [13127.4 to 20932.0]
  Anti-HPV-16, Month 24: number analyzed (Participants) | 87
  Anti-HPV-16, Month 24 | 10003.7 [8114.1 to 12333.4]
  Anti-HPV-16, Month 36 | 9214.3 [7112.3 to 11937.5]
  Anti-HPV-18, Day 0 | 20.0 [20.0 to 20.0]
  Anti-HPV-18, Month 13 | 39994.7 [33327.2 to 47996.1]
  Anti-HPV-18, Month 18 | 9495.4 [7744.4 to 11642.2]
  Anti-HPV-18, Month 24: number analyzed (Participants) | 87
  Anti-HPV-18, Month 24 | 5464.1 [4377.8 to 6819.8]
  Anti-HPV-18, Month 36 | 4046.4 [3278.0 to 4994.8]

8. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Titers (by PBNA) in a Subset of Subjects From Cervarix 1 Group and Cervarix 2 Group
Description: Antibody titers were expressed as GMTs. The cut-off of the assay was 40 ED50 for both anti-HPV-16 and anti-HPV-18. The assay was performed on a subset of 100 subjects per study group.
Time Frame: At Day 0 and at Months 7, 12, 18, 24 and 36
Population: The analysis was based on the Month 36 ATP cohort for immunogenicity which included a subset of 100 subjects per study group, who returned for blood sampling at Month 36 and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination at the specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix 1 Group | Cervarix 2 Group
Number analyzed (Participants) | 96 | 92
Titers
  Anti-HPV-16, Day 0 | 21.3 [18.8 to 24.2] | 23.5 [20.7 to 26.6]
  Anti-HPV-16, Month 7 | 82975.9 [67377.4 to 102185.6] | 31407.6 [24181.5 to 40793.0]
  Anti-HPV-16, Month 12 | 14872.1 [12025.5 to 18392.4] | 15801.8 [12069.8 to 20687.8]
  Anti-HPV-16, Month 18: number analyzed (Participants) | 95 | 92
  Anti-HPV-16, Month 18 | 7393.6 [5986.6 to 9131.1] | 8246.4 [6224.6 to 10925.0]
  Anti-HPV-16, Month 24 | 6216.5 [5111.0 to 7561.1] | 7267.5 [5423.4 to 9738.6]
  Anti-HPV-16, Month 36 | 7762.7 [6218.6 to 9690.1] | 5063.7 [3800.4 to 6746.9]
  Anti-HPV-18, Day 0 | 21.0 [19.0 to 23.5] | 22.4 [20.4 to 24.5]
  Anti-HPV-18, Month 7 | 24833.1 [20777.0 to 29681.1] | 13935.6 [10991.0 to 17669.0]
  Anti-HPV-18, Month 12 | 5914.5 [4756.0 to 7355.4] | 5066.5 [3818.9 to 6721.7]
  Anti-HPV-18, Month 18: number analyzed (Participants) | 95 | 92
  Anti-HPV-18, Month 18 | 3961.2 [3153.8 to 4975.4] | 2958.2 [2213.9 to 3952.6]
  Anti-HPV-18, Month 24 | 2849.4 [2276.0 to 3567.2] | 2524.3 [1860.4 to 3425.2]
  Anti-HPV-18, Month 36: number analyzed (Participants) | 95 | 92
  Anti-HPV-18, Month 36 | 2416.4 [1905.9 to 3063.5] | 1956.2 [1488.5 to 2570.7]

9. Secondary Outcome: Cell-mediated Immunogenicity Related to Anti-HPV-16 Specific T Cell-mediated Immune Response (CMI) for Cervarix 1 Group and Cervarix 2 Group in a Sub-cohort of Subjects
Description: The CMI response represents the measure of the cytokines production [i.e. interleukin-2 (IL-2), interferon gamma (IFN-γ), tumor necrosis factor alpha (TNF-α) and the cluster of differentiation 40 Ligand (CD40L)] by HPV-antigen specific T lymphocytes and measured by intracellular cytokine staining (ICS) assay for HPV-16. The frequency was presented as number of cytokine-positive cluster of differentiation (CD)4 i.e. CD4+/CD8+ cells per million CD4+/CD8+ cells. All doubles = T cell expressing at least 2 cytokines. Results were tabulated by the pre-vaccination status of the subjects, where S- = seronegative subjects (antibody concentration < cut-off value) prior to vaccination. S+ = seropositive subjects (antibody concentration ≥ cut-off value) prior to vaccination. The assay was performed on a subset of 100 subjects per study group.
Time Frame: At Day 0 and at Months 7, 12, 24 and 36
Population: The analysis was based on the Month 36 ATP cohort for immunogenicity which included a sub-cohort of 100 subjects per study group, who returned for blood sampling at Month 36 and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination at the specified time points.
Measure: Median (Inter-Quartile Range); unit: cells/million T cells
Arm/Group | Cervarix 1 Group | Cervarix 2 Group
Number analyzed (Participants) | 84 | 70
cells/million T cells
  Anti-HPV-16, CD4 all doubles, S-, Day 0: number analyzed (Participants) | 81 | 68
  Anti-HPV-16, CD4 all doubles, S-, Day 0 | 88.0 [62.0 to 152.0] | 120.0 [67.0 to 185.5]
  Anti-HPV-16, CD4 all doubles, S-, Month 7: number analyzed (Participants) | 69 | 50
  Anti-HPV-16, CD4 all doubles, S-, Month 7 | 3953.0 [1866.0 to 7025.0] | 3426.0 [1889.0 to 5214.0]
  Anti-HPV-16, CD4 all doubles, S-, Month 12 | 2491.0 [1387.5 to 5543.5] | 2278.5 [1225.0 to 3363.0]
  Anti-HPV-16, CD4 all doubles, S-, Month 24: number analyzed (Participants) | 78 | 67
  Anti-HPV-16, CD4 all doubles, S-, Month 24 | 2698.0 [1231.0 to 5147.0] | 2401.0 [1231.0 to 3641.0]
  Anti-HPV-16, CD4 all doubles, S-, Month 36: number analyzed (Participants) | 75 | 57
  Anti-HPV-16, CD4 all doubles, S-, Month 36 | 1951.0 [1085.0 to 5130.0] | 2073.0 [1012.0 to 2836.0]
  Anti-HPV-16, CD4 all doubles, S+, Day 0: number analyzed (Participants) | 8 | 14
  Anti-HPV-16, CD4 all doubles, S+, Day 0 | 77.5 [57.0 to 192.0] | 100.0 [60.0 to 269.0]
  Anti-HPV-16, CD4 all doubles, S+, Month 7: number analyzed (Participants) | 8 | 13
  Anti-HPV-16, CD4 all doubles, S+, Month 7 | 5019.5 [1353.0 to 7343.0] | 1820.0 [1311.0 to 3021.0]
  Anti-HPV-16, CD4 all doubles, S+, Month 12: number analyzed (Participants) | 9 | 14
  Anti-HPV-16, CD4 all doubles, S+, Month 12 | 2603.0 [1003.0 to 3350.0] | 1423.5 [876.0 to 3747.0]
  Anti-HPV-16, CD4 all doubles, S+, Month 24: number analyzed (Participants) | 9 | 12
  Anti-HPV-16, CD4 all doubles, S+, Month 24 | 2552.0 [1156.0 to 3963.0] | 1404.0 [1050.0 to 2856.5]
  Anti-HPV-16, CD4 all doubles, S+, Month 36: number analyzed (Participants) | 7 | 12
  Anti-HPV-16, CD4 all doubles, S+, Month 36 | 2180.0 [1293.0 to 3383.0] | 1310.0 [939.0 to 2614.5]
  Anti-HPV-16, CD4-d-CD40L, S-, Day 0: number analyzed (Participants) | 81 | 68
  Anti-HPV-16, CD4-d-CD40L, S-, Day 0 | 70.0 [42.0 to 130.0] | 97.0 [49.0 to 144.0]
  Anti-HPV-16, CD4-d-CD40L, S-, Month 7: number analyzed (Participants) | 69 | 50
  Anti-HPV-16, CD4-d-CD40L, S-, Month 7 | 3531.0 [1676.0 to 6528.0] | 3196.0 [1692.0 to 4771.0]
  Anti-HPV-16, CD4-d-CD40L, S-, Month 12 | 2439.5 [1342.5 to 5376.0] | 2255.5 [1185.0 to 3290.0]
  Anti-HPV-16, CD4-d-CD40L, S-, Month 24: number analyzed (Participants) | 78 | 67
  Anti-HPV-16, CD4-d-CD40L, S-, Month 24 | 2443.0 [1111.0 to 4922.0] | 2344.0 [1031.0 to 3323.0]
  Anti-HPV-16, CD4-d-CD40L, S-, Month 36: number analyzed (Participants) | 75 | 57
  Anti-HPV-16, CD4-d-CD40L, S-, Month 36 | 1935.0 [1048.0 to 5061.0] | 2027.0 [978.0 to 2806.0]
  Anti-HPV-16, CD4-d-CD40L, S+, Day 0: number analyzed (Participants) | 8 | 14
  Anti-HPV-16, CD4-d-CD40L, S+, Day 0 | 57.5 [39.5 to 162.0] | 72.5 [40.0 to 186.0]
  Anti-HPV-16, CD4-d-CD40L, S+, Month 7: number analyzed (Participants) | 8 | 13
  Anti-HPV-16, CD4-d-CD40L, S+, Month 7 | 4979.5 [1290.5 to 7001.5] | 1655.0 [1050.0 to 2440.0]
  Anti-HPV-16, CD4-d-CD40L, S+, Month 12: number analyzed (Participants) | 9 | 14
  Anti-HPV-16, CD4-d-CD40L, S+, Month 12 | 2587.0 [975.0 to 3305.0] | 1412.5 [832.0 to 3677.0]
  Anti-HPV-16, CD4-d-CD40L, S+, Month 24: number analyzed (Participants) | 9 | 12
  Anti-HPV-16, CD4-d-CD40L, S+, Month 24 | 2456.0 [945.0 to 3931.0] | 1285.0 [962.5 to 1953.5]
  Anti-HPV-16, CD4-d-CD40L, S+, Month 36: number analyzed (Participants) | 7 | 12
  Anti-HPV-16, CD4-d-CD40L, S+, Month 36 | 2109.0 [1178.0 to 3343.0] | 1279.0 [928.0 to 2496.5]
  Anti-HPV-16, CD4-d-IFNγ, S-, Day 0: number analyzed (Participants) | 81 | 68
  Anti-HPV-16, CD4-d-IFNγ, S-, Day 0 | 44.0 [19.0 to 67.0] | 39.5 [19.5 to 72.0]
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 7: number analyzed (Participants) | 69 | 50
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 7 | 840.0 [503.0 to 1538.0] | 657.0 [474.0 to 1185.0]
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 12 | 546.0 [176.5 to 1007.5] | 362.0 [202.0 to 644.0]
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 24: number analyzed (Participants) | 78 | 67
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 24 | 644.5 [294.0 to 1318.0] | 449.0 [204.0 to 884.0]
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 36: number analyzed (Participants) | 75 | 57
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 36 | 562.0 [273.0 to 1334.0] | 391.0 [215.0 to 824.0]
  Anti-HPV-16, CD4-d-IFNγ, S+, Day 0: number analyzed (Participants) | 8 | 14
  Anti-HPV-16, CD4-d-IFNγ, S+, Day 0 | 38.5 [26.5 to 86.0] | 50.5 [31.0 to 75.0]
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 7: number analyzed (Participants) | 8 | 13
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 7 | 881.5 [462.5 to 2704.0] | 489.0 [244.0 to 814.0]
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 12: number analyzed (Participants) | 9 | 14
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 12 | 533.0 [336.0 to 827.0] | 329.0 [183.0 to 481.0]
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 24: number analyzed (Participants) | 9 | 12
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 24 | 579.0 [398.0 to 897.0] | 310.5 [221.5 to 595.5]
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 36: number analyzed (Participants) | 7 | 12
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 36 | 651.0 [520.0 to 998.0] | 564.0 [185.5 to 714.5]
  Anti-HPV-16, CD4-d-IL-2, S-, Day 0: number analyzed (Participants) | 81 | 68
  Anti-HPV-16, CD4-d-IL-2, S-, Day 0 | 59.0 [35.0 to 103.0] | 85.5 [43.5 to 143.0]
  Anti-HPV-16, CD4-d-IL-2, S-, Month 7: number analyzed (Participants) | 69 | 50
  Anti-HPV-16, CD4-d-IL-2, S-, Month 7 | 3808.0 [1728.0 to 6787.0] | 3212.5 [1788.0 to 5010.0]
  Anti-HPV-16, CD4-d-IL-2, S-, Month 12 | 2402.5 [1308.5 to 5242.0] | 2184.5 [1156.0 to 3238.0]
  Anti-HPV-16, CD4-d-IL-2, S-, Month 24: number analyzed (Participants) | 78 | 67
  Anti-HPV-16, CD4-d-IL-2, S-, Month 24 | 2477.0 [1140.0 to 4680.0] | 2282.0 [1138.0 to 3392.0]
  Anti-HPV-16, CD4-d-IL-2, S-, Month 36: number analyzed (Participants) | 75 | 57
  Anti-HPV-16, CD4-d-IL-2, S-, Month 36 | 1881.0 [958.0 to 4912.0] | 1922.0 [892.0 to 2708.0]
  Anti-HPV-16, CD4-d-IL-2, S+, Day 0: number analyzed (Participants) | 8 | 14
  Anti-HPV-16, CD4-d-IL-2, S+, Day 0 | 68.0 [23.0 to 147.5] | 77.5 [39.0 to 229.0]
  Anti-HPV-16, CD4-d-IL-2, S+, Month 7: number analyzed (Participants) | 8 | 13
  Anti-HPV-16, CD4-d-IL-2, S+, Month 7 | 4886.0 [1162.5 to 6906.0] | 1573.0 [1202.0 to 2924.0]
  Anti-HPV-16, CD4-d-IL-2, S+, Month 12: number analyzed (Participants) | 9 | 14
  Anti-HPV-16, CD4-d-IL-2, S+, Month 12 | 2339.0 [877.0 to 3166.0] | 1372.0 [868.0 to 3692.0]
  Anti-HPV-16, CD4-d-IL-2, S+, Month 24: number analyzed (Participants) | 9 | 12
  Anti-HPV-16, CD4-d-IL-2, S+, Month 24 | 2454.0 [1026.0 to 3931.0] | 1226.5 [969.0 to 2392.5]
  Anti-HPV-16, CD4-d-IL-2, S+, Month 36: number analyzed (Participants) | 7 | 12
  Anti-HPV-16, CD4-d-IL-2, S+, Month 36 | 2135.0 [1221.0 to 3291.0] | 1243.0 [910.5 to 2382.5]
  Anti-HPV-16, CD4-d-TNFα, S-, Day 0: number analyzed (Participants) | 81 | 68
  Anti-HPV-16, CD4-d-TNFα, S-, Day 0 | 59.0 [37.0 to 93.0] | 68.0 [29.5 to 110.5]
  Anti-HPV-16, CD4-d-TNFα, S-, Month 7: number analyzed (Participants) | 69 | 50
  Anti-HPV-16, CD4-d-TNFα, S-, Month 7 | 2474.0 [1311.0 to 4800.0] | 2575.5 [1224.0 to 3675.0]
  Anti-HPV-16, CD4-d-TNFα, S-, Month 12 | 1944.0 [814.5 to 4150.0] | 1726.0 [919.0 to 2481.0]
  Anti-HPV-16, CD4-d-TNFα, S-, Month 24: number analyzed (Participants) | 78 | 67
  Anti-HPV-16, CD4-d-TNFα, S-, Month 24 | 2181.5 [886.0 to 4177.0] | 1970.0 [773.0 to 2758.0]
  Anti-HPV-16, CD4-d-TNFα, S-, Month 36: number analyzed (Participants) | 75 | 57
  Anti-HPV-16, CD4-d-TNFα, S-, Month 36 | 1595.0 [700.0 to 3836.0] | 1390.0 [672.0 to 2092.0]
  Anti-HPV-16, CD4-d-TNFα, S+, Day 0: number analyzed (Participants) | 8 | 14
  Anti-HPV-16, CD4-d-TNFα, S+, Day 0 | 47.0 [32.0 to 131.0] | 64.0 [49.0 to 120.0]
  Anti-HPV-16, CD4-d-TNFα, S+, Month 7: number analyzed (Participants) | 8 | 13
  Anti-HPV-16, CD4-d-TNFα, S+, Month 7 | 2058.5 [1047.0 to 3933.0] | 1273.0 [949.0 to 2372.0]
  Anti-HPV-16, CD4-d-TNFα, S+, Month 12: number analyzed (Participants) | 9 | 14
  Anti-HPV-16, CD4-d-TNFα, S+, Month 12 | 1826.0 [875.0 to 2703.0] | 1171.0 [733.0 to 2828.0]
  Anti-HPV-16, CD4-d-TNFα, S+, Month 24: number analyzed (Participants) | 9 | 12
  Anti-HPV-16, CD4-d-TNFα, S+, Month 24 | 1851.0 [1039.0 to 2259.0] | 1061.5 [878.5 to 2421.5]
  Anti-HPV-16, CD4-d-TNFα, S+, Month 36: number analyzed (Participants) | 7 | 12
  Anti-HPV-16, CD4-d-TNFα, S+, Month 36 | 1138.0 [1031.0 to 2506.0] | 1057.0 [732.0 to 2009.0]
  Anti-HPV-16, CD8-all doubles, S-, Day 0: number analyzed (Participants) | 81 | 68
  Anti-HPV-16, CD8-all doubles, S-, Day 0 | 11.0 [11.0 to 41.0] | 11.0 [11.0 to 44.0]
  Anti-HPV-16, CD8-all doubles, S-, Month 7: number analyzed (Participants) | 69 | 50
  Anti-HPV-16, CD8-all doubles, S-, Month 7 | 11.0 [11.0 to 41.0] | 11.0 [11.0 to 36.0]
  Anti-HPV-16, CD8 all doubles, S-, Month 12 | 30.5 [11.0 to 45.5] | 29.5 [11.0 to 50.0]
  Anti-HPV-16, CD8-all doubles, S-, Month 24: number analyzed (Participants) | 78 | 67
  Anti-HPV-16, CD8-all doubles, S-, Month 24 | 11.0 [11.0 to 53.0] | 11.0 [11.0 to 54.0]
  Anti-HPV-16, CD8-all doubles, S-, Month 36: number analyzed (Participants) | 75 | 57
  Anti-HPV-16, CD8-all doubles, S-, Month 36 | 37.0 [11.0 to 72.0] | 35.0 [11.0 to 59.0]
  Anti-HPV-16, CD8-all doubles, S+, Day 0: number analyzed (Participants) | 8 | 14
  Anti-HPV-16, CD8-all doubles, S+, Day 0 | 11.0 [11.0 to 49.0] | 35.5 [26.0 to 41.0]
  Anti-HPV-16, CD8-all doubles, S+, Month 7: number analyzed (Participants) | 8 | 13
  Anti-HPV-16, CD8-all doubles, S+, Month 7 | 11.0 [11.0 to 30.5] | 33.0 [11.0 to 43.0]
  Anti-HPV-16, CD8 all doubles, S+, Month 12: number analyzed (Participants) | 9 | 14
  Anti-HPV-16, CD8 all doubles, S+, Month 12 | 52.0 [49.0 to 77.0] | 29.0 [11.0 to 57.0]
  Anti-HPV-16, CD8-all doubles, S+, Month 24: number analyzed (Participants) | 9 | 12
  Anti-HPV-16, CD8-all doubles, S+, Month 24 | 49.0 [12.0 to 63.0] | 11.0 [11.0 to 56.0]
  Anti-HPV-16, CD8-all doubles, S+, Month 36: number analyzed (Participants) | 7 | 12
  Anti-HPV-16, CD8-all doubles, S+, Month 36 | 27.0 [11.0 to 123.0] | 11.0 [11.0 to 49.0]
  Anti-HPV-16, CD8-d-CD40L, S-, Day 0: number analyzed (Participants) | 81 | 68
  Anti-HPV-16, CD8-d-CD40L, S-, Day 0 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-CD40L, S-, Month 7: number analyzed (Participants) | 69 | 50
  Anti-HPV-16, CD8-d-CD40L, S-, Month 7 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-CD40L, S-, Month 12 | 7.0 [7.0 to 32.0] | 7.0 [7.0 to 37.0]
  Anti-HPV-16, CD8-d-CD40L, S-, Month 24: number analyzed (Participants) | 78 | 67
  Anti-HPV-16, CD8-d-CD40L, S-, Month 24 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 31.0]
  Anti-HPV-16, CD8-d-CD40L, S-, Month 36: number analyzed (Participants) | 75 | 57
  Anti-HPV-16, CD8-d-CD40L, S-, Month 36 | 11.0 [7.0 to 52.0] | 7.0 [7.0 to 32.0]
  Anti-HPV-16, CD8-d-CD40L, S+, Day 0: number analyzed (Participants) | 8 | 14
  Anti-HPV-16, CD8-d-CD40L, S+, Day 0 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-CD40L, S+, Month 7: number analyzed (Participants) | 8 | 13
  Anti-HPV-16, CD8-d-CD40L, S+, Month 7 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 22.0]
  Anti-HPV-16, CD8-d-CD40L, S+, Month 12: number analyzed (Participants) | 9 | 14
  Anti-HPV-16, CD8-d-CD40L, S+, Month 12 | 45.0 [7.0 to 48.0] | 15.0 [7.0 to 37.0]
  Anti-HPV-16, CD8-d-CD40L, S+, Month 24: number analyzed (Participants) | 9 | 12
  Anti-HPV-16, CD8-d-CD40L, S+, Month 24 | 7.0 [7.0 to 46.0] | 7.0 [7.0 to 17.0]
  Anti-HPV-16, CD8-d-CD40L, S+, Month 36: number analyzed (Participants) | 7 | 12
  Anti-HPV-16, CD8-d-CD40L, S+, Month 36 | 7.0 [7.0 to 27.0] | 7.0 [7.0 to 15.0]
  Anti-HPV-16, CD8-d-IFNγ, S-, Day 0: number analyzed (Participants) | 81 | 68
  Anti-HPV-16, CD8-d-IFNγ, S-, Day 0 | 7.0 [7.0 to 32.0] | 7.0 [7.0 to 37.0]
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 7: number analyzed (Participants) | 69 | 50
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 7 | 7.0 [7.0 to 35.0] | 7.0 [7.0 to 26.0]
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 12 | 7.0 [7.0 to 38.0] | 7.0 [7.0 to 46.0]
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 24: number analyzed (Participants) | 78 | 67
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 24 | 7.0 [7.0 to 37.0] | 7.0 [7.0 to 42.0]
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 36: number analyzed (Participants) | 75 | 57
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 36 | 11.0 [7.0 to 44.0] | 25.0 [7.0 to 44.0]
  Anti-HPV-16, CD8-d-IFNγ, S+, Day 0: number analyzed (Participants) | 8 | 14
  Anti-HPV-16, CD8-d-IFNγ, S+, Day 0 | 7.0 [7.0 to 45.0] | 31.5 [22.0 to 37.0]
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 7: number analyzed (Participants) | 8 | 13
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 7 | 7.0 [7.0 to 7.0] | 22.0 [7.0 to 30.0]
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 12: number analyzed (Participants) | 9 | 14
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 12 | 46.0 [31.0 to 54.0] | 15.0 [7.0 to 40.0]
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 24: number analyzed (Participants) | 9 | 12
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 24 | 8.0 [7.0 to 46.0] | 7.0 [7.0 to 23.0]
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 36: number analyzed (Participants) | 7 | 12
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 36 | 7.0 [7.0 to 63.0] | 7.0 [7.0 to 45.0]
  Anti-HPV-16, CD8-d-IL-2, S-, Day 0: number analyzed (Participants) | 81 | 68
  Anti-HPV-16, CD8-d-IL-2, S-, Day 0 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-IL-2, S-, Month 7: number analyzed (Participants) | 69 | 50
  Anti-HPV-16, CD8-d-IL-2, S-, Month 7 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-IL-2, S-, Month 12 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-IL-2, S-, Month 24: number analyzed (Participants) | 78 | 67
  Anti-HPV-16, CD8-d-IL-2, S-, Month 24 | 7.0 [7.0 to 30.0] | 7.0 [7.0 to 30.0]
  Anti-HPV-16, CD8-d-IL-2, S-, Month 36: number analyzed (Participants) | 75 | 57
  Anti-HPV-16, CD8-d-IL-2, S-, Month 36 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-IL-2, S+, Day 0: number analyzed (Participants) | 8 | 14
  Anti-HPV-16, CD8-d-IL-2, S+, Day 0 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-IL-2, S+, Month 7: number analyzed (Participants) | 8 | 13
  Anti-HPV-16, CD8-d-IL-2, S+, Month 7 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 28.0]
  Anti-HPV-16, CD8-d-IL-2, S+, Month 12: number analyzed (Participants) | 9 | 14
  Anti-HPV-16, CD8-d-IL-2, S+, Month 12 | 7.0 [7.0 to 31.0] | 7.0 [7.0 to 23.0]
  Anti-HPV-16, CD8-d-IL-2, S+, Month 24: number analyzed (Participants) | 9 | 12
  Anti-HPV-16, CD8-d-IL-2, S+, Month 24 | 7.0 [7.0 to 45.0] | 7.0 [7.0 to 13.0]
  Anti-HPV-16, CD8-d-IL-2, S+, Month 36: number analyzed (Participants) | 7 | 12
  Anti-HPV-16, CD8-d-IL-2, S+, Month 36 | 7 [7.0 to 23.0] | 7 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-TNFα, S-, Day 0: number analyzed (Participants) | 81 | 68
  Anti-HPV-16, CD8-d-TNFα, S-, Day 0 | 7.0 [7.0 to 29.0] | 7.0 [7.0 to 28.5]
  Anti-HPV-16, CD8-d-TNFα, S-, Month 7: number analyzed (Participants) | 69 | 50
  Anti-HPV-16, CD8-d-TNFα, S-, Month 7 | 7.0 [7.0 to 33.0] | 7.0 [7.0 to 32.0]
  Anti-HPV-16, CD8-d-TNFα, S-, Month 12 | 7.0 [7.0 to 38.0] | 7.0 [7.0 to 33.0]
  Anti-HPV-16, CD8-d-TNFα, S-, Month 24: number analyzed (Participants) | 78 | 67
  Anti-HPV-16, CD8-d-TNFα, S-, Month 24 | 7.0 [7.0 to 37.0] | 7.0 [7.0 to 24.0]
  Anti-HPV-16, CD8-d-TNFα, S-, Month 36: number analyzed (Participants) | 75 | 57
  Anti-HPV-16, CD8-d-TNFα, S-, Month 36 | 7 [7.0 to 36.0] | 7 [7.0 to 32.0]
  Anti-HPV-16, CD8-d-TNFα, S+, Day 0: number analyzed (Participants) | 8 | 14
  Anti-HPV-16, CD8-d-TNFα, S+, Day 0 | 7.0 [7.0 to 30.5] | 14.5 [7.0 to 31.0]
  Anti-HPV-16, CD8-d-TNFα, S+, Month 7: number analyzed (Participants) | 8 | 13
  Anti-HPV-16, CD8-d-TNFα, S+, Month 7 | 7.0 [7.0 to 26.5] | 22.0 [7.0 to 30.0]
  Anti-HPV-16, CD8-d-TNFα, S+, Month 12: number analyzed (Participants) | 9 | 14
  Anti-HPV-16, CD8-d-TNFα, S+, Month 12 | 8.0 [7.0 to 54.0] | 23.0 [7.0 to 30.0]
  Anti-HPV-16, CD8-d-TNFα, S+, Month 24: number analyzed (Participants) | 9 | 12
  Anti-HPV-16, CD8-d-TNFα, S+, Month 24 | 8.0 [7.0 to 42.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-TNFα, S+, Month 36: number analyzed (Participants) | 7 | 12
  Anti-HPV-16, CD8-d-TNFα, S+, Month 36 | 7.0 [7.0 to 119.0] | 7.0 [7.0 to 7.0]

10. Secondary Outcome: Cell-mediated Immunogenicity Related to Anti-HPV-18 Specific T CMI Response for Cervarix 1 Group and Cervarix 2 Group in a Sub-cohort of Subjects
Description: The CMI response represents the measure of the cytokines production [IL-2, IFN-γ, TNF-α, and CD40L] by HPV-antigen specific T lymphocytes and measured by ICS assay for HPV-18. The frequency was presented as a number of cytokine-producing CD4+/CD8+ cells per million CD4+/CD8+ cells. All doubles = T cell expressing at least 2 cytokines. Results were tabulated by the pre-vaccination status of the subjects, where S- = seronegative subjects (antibody concentration < the cut-off value) prior to vaccination. S+ = seropositive subjects (antibody concentration ≥ cut-off value) prior to vaccination. The assay was performed on a subset of 100 subjects per study group.
Time Frame: At Day 0 and at Months 7, 12, 24 and 36
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: cells/million T cells
Arm/Group | Cervarix 1 Group | Cervarix 2 Group
Number analyzed (Participants) | 83 | 72
cells/million T cells
  Anti-HPV-18, CD4 all doubles, S-, Day 0: number analyzed (Participants) | 77 | 69
  Anti-HPV-18, CD4 all doubles, S-, Day 0 | 86.0 [61.0 to 129.0] | 112.0 [75.0 to 177.0]
  Anti-HPV-18, CD4 all doubles, S-, Month 7: number analyzed (Participants) | 65 | 53
  Anti-HPV-18, CD4 all doubles, S-, Month 7 | 2780.0 [1606.0 to 4289.0] | 1864.0 [1158.0 to 2565.0]
  Anti-HPV-18, CD4 all doubles, S-, Month 12 | 2039.0 [1053.0 to 3481.0] | 1246.5 [814.0 to 2045.5]
  Anti-HPV-18, CD4 all doubles, S-, Month 24: number analyzed (Participants) | 76 | 68
  Anti-HPV-18, CD4 all doubles, S-, Month 24 | 1815.5 [877.5 to 3193.0] | 1355.0 [638.5 to 2106.0]
  Anti-HPV-18, CD4 all doubles, S-, Month 36: number analyzed (Participants) | 72 | 56
  Anti-HPV-18, CD4 all doubles, S-, Month 36 | 1609.0 [716.0 to 3322.0] | 1246.0 [676.5 to 1751.0]
  Anti-HPV-18, CD4 all doubles, S+, Day 0: number analyzed (Participants) | 11 | 14
  Anti-HPV-18, CD4 all doubles, S+, Day 0 | 125.0 [61.0 to 227.0] | 128.0 [71.0 to 153.0]
  Anti-HPV-18, CD4 all doubles, S+, Month 7: number analyzed (Participants) | 11 | 11
  Anti-HPV-18, CD4 all doubles, S+, Month 7 | 1593.0 [786.0 to 4012.0] | 1498.0 [808.0 to 2727.0]
  Anti-HPV-18, CD4 all doubles, S+, Month 12: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD4 all doubles, S+, Month 12 | 868.0 [576.0 to 2069.0] | 787.0 [597.0 to 1771.0]
  Anti-HPV-18, CD4 all doubles, S+, Month 24: number analyzed (Participants) | 10 | 12
  Anti-HPV-18, CD4 all doubles, S+, Month 24 | 710.5 [523.0 to 2329.0] | 885.0 [475.5 to 2147.5]
  Anti-HPV-18, CD4 all doubles, S+, Month 36: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD4 all doubles, S+, Month 36 | 808.5 [624.0 to 1764.0] | 598.0 [367.0 to 1414.0]
  Anti-HPV-18, CD4-d-CD40L, S-, Day 0: number analyzed (Participants) | 77 | 69
  Anti-HPV-18, CD4-d-CD40L, S-, Day 0 | 62.0 [35.0 to 105.0] | 88.0 [49.0 to 155.0]
  Anti-HPV-18, CD4-d-CD40L, S-, Month 7: number analyzed (Participants) | 65 | 53
  Anti-HPV-18, CD4-d-CD40L, S-, Month 7 | 2634.0 [1331.0 to 3748.0] | 1700.0 [993.0 to 2324.0]
  Anti-HPV-18, CD4-d-CD40L, S-, Month 12 | 1967.0 [1019.0 to 3362.0] | 1206.5 [797.5 to 2006.0]
  Anti-HPV-18, CD4-d-CD40L, S-, Month 24: number analyzed (Participants) | 76 | 68
  Anti-HPV-18, CD4-d-CD40L, S-, Month 24 | 1632.0 [807.0 to 3133.0] | 1290.5 [600.5 to 1911.0]
  Anti-HPV-18, CD4-d-CD40L, S-, Month 36: number analyzed (Participants) | 72 | 56
  Anti-HPV-18, CD4-d-CD40L, S-, Month 36 | 1543.0 [686.0 to 3258.0] | 1222.0 [670.0 to 1665.0]
  Anti-HPV-18, CD4-d-CD40L, S+, Day 0: number analyzed (Participants) | 11 | 14
  Anti-HPV-18, CD4-d-CD40L, S+, Day 0 | 121.0 [50.0 to 223.0] | 110.5 [44.0 to 142.0]
  Anti-HPV-18, CD4-d-CD40L, S+, Month 7: number analyzed (Participants) | 11 | 11
  Anti-HPV-18, CD4-d-CD40L, S+, Month 7 | 1419.0 [729.0 to 3704.0] | 1377.0 [703.0 to 2511.0]
  Anti-HPV-18, CD4-d-CD40L, S+, Month 12: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD4-d-CD40L, S+, Month 12 | 830.0 [572.0 to 2008.0] | 767.0 [539.0 to 1724.0]
  Anti-HPV-18, CD4-d-CD40L, S+, Month 24: number analyzed (Participants) | 10 | 12
  Anti-HPV-18, CD4-d-CD40L, S+, Month 24 | 652.0 [475.0 to 2151.0] | 867.0 [431.0 to 1963.5]
  Anti-HPV-18, CD4-d-CD40L, S+, Month 36: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD4-d-CD40L, S+, Month 36 | 794.0 [604.0 to 1721.0] | 594.0 [350.0 to 1356.0]
  Anti-HPV-18, CD4-d-IFNγ, S-, Day 0: number analyzed (Participants) | 77 | 69
  Anti-HPV-18, CD4-d-IFNγ, S-, Day 0 | 32.0 [19.0 to 55.0] | 32.0 [19.0 to 68.0]
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 7: number analyzed (Participants) | 65 | 53
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 7 | 562.0 [220.0 to 952.0] | 350.0 [192.0 to 554.0]
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 12 | 354.0 [132.0 to 669.0] | 216.5 [111.5 to 390.0]
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 24: number analyzed (Participants) | 76 | 68
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 24 | 326.5 [166.5 to 799.5] | 205.5 [108.5 to 538.0]
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 36: number analyzed (Participants) | 72 | 56
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 36 | 304.5 [168.5 to 757.0] | 233.5 [114.5 to 485.5]
  Anti-HPV-18, CD4-d-IFNγ, S+, Day 0: number analyzed (Participants) | 11 | 14
  Anti-HPV-18, CD4-d-IFNγ, S+, Day 0 | 55.0 [19.0 to 70.0] | 28.0 [19.0 to 48.0]
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 7: number analyzed (Participants) | 11 | 11
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 7 | 628.0 [186.0 to 1186.0] | 376.0 [234.0 to 580.0]
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 12: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 12 | 244.5 [120.0 to 535.0] | 161.0 [85.0 to 344.0]
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 24: number analyzed (Participants) | 10 | 12
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 24 | 295.5 [108.0 to 636.0] | 270.5 [94.5 to 455.5]
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 36: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 36 | 356.0 [278.0 to 417.0] | 239.0 [102.0 to 422.0]
  Anti-HPV-18, CD4-d-IL-2, S-, Day 0: number analyzed (Participants) | 77 | 69
  Anti-HPV-18, CD4-d-IL-2, S-, Day 0 | 57.0 [30.0 to 96.0] | 81.0 [36.0 to 127.0]
  Anti-HPV-18, CD4-d-IL-2, S-, Month 7: number analyzed (Participants) | 65 | 53
  Anti-HPV-18, CD4-d-IL-2, S-, Month 7 | 2611.0 [1452.0 to 3953.0] | 1725.0 [1026.0 to 2329.0]
  Anti-HPV-18, CD4-d-IL-2, S-, Month 12 | 1959.0 [1009.0 to 3269.0] | 1172.5 [755.5 to 1916.0]
  Anti-HPV-18, CD4-d-IL-2, S-, Month 24: number analyzed (Participants) | 76 | 68
  Anti-HPV-18, CD4-d-IL-2, S-, Month 24 | 1638.5 [851.5 to 3084.0] | 1306.0 [589.0 to 1977.5]
  Anti-HPV-18, CD4-d-IL-2, S-, Month 36: number analyzed (Participants) | 72 | 56
  Anti-HPV-18, CD4-d-IL-2, S-, Month 36 | 1495.0 [661.0 to 3065.0] | 1183.5 [586.5 to 1684.5]
  Anti-HPV-18, CD4-d-IL-2, S+, Day 0: number analyzed (Participants) | 11 | 14
  Anti-HPV-18, CD4-d-IL-2, S+, Day 0 | 65.0 [31.0 to 137.0] | 96.5 [48.0 to 102.0]
  Anti-HPV-18, CD4-d-IL-2, S+, Month 7: number analyzed (Participants) | 11 | 11
  Anti-HPV-18, CD4-d-IL-2, S+, Month 7 | 1470.0 [691.0 to 3887.0] | 1231.0 [690.0 to 2313.0]
  Anti-HPV-18, CD4-d-IL-2, S+, Month 12: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD4-d-IL-2, S+, Month 12 | 847.5 [556.0 to 2022.0] | 783.0 [514.0 to 1650.0]
  Anti-HPV-18, CD4-d-IL-2, S+, Month 24: number analyzed (Participants) | 10 | 12
  Anti-HPV-18, CD4-d-IL-2, S+, Month 24 | 652.5 [448.0 to 2269.0] | 705.5 [433.0 to 2041.5]
  Anti-HPV-18, CD4-d-IL-2, S+, Month 36: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD4-d-IL-2, S+, Month 36 | 777.0 [589.0 to 1669.0] | 554.0 [333.0 to 1370.0]
  Anti-HPV-18, CD4-d-TNFα, S-, Day 0: number analyzed (Participants) | 77 | 69
  Anti-HPV-18, CD4-d-TNFα, S-, Day 0 | 49.0 [31.0 to 72.0] | 73.0 [27.0 to 138.0]
  Anti-HPV-18, CD4-d-TNFα, S-, Month 7: number analyzed (Participants) | 65 | 53
  Anti-HPV-18, CD4-d-TNFα, S-, Month 7 | 1699.0 [979.0 to 2832.0] | 1394.0 [824.0 to 2060.0]
  Anti-HPV-18, CD4-d-TNFα, S-, Month 12 | 1573.0 [715.0 to 2662.0] | 991.0 [599.0 to 1617.0]
  Anti-HPV-18, CD4-d-TNFα, S-, Month 24: number analyzed (Participants) | 76 | 68
  Anti-HPV-18, CD4-d-TNFα, S-, Month 24 | 1434.0 [637.5 to 2506.0] | 1102.5 [543.0 to 1580.0]
  Anti-HPV-18, CD4-d-TNFα, S-, Month 36: number analyzed (Participants) | 72 | 56
  Anti-HPV-18, CD4-d-TNFα, S-, Month 36 | 1268.0 [473.5 to 2130.0] | 868.5 [520.0 to 1296.5]
  Anti-HPV-18, CD4-d-TNFα, S+, Day 0: number analyzed (Participants) | 11 | 14
  Anti-HPV-18, CD4-d-TNFα, S+, Day 0 | 51.0 [44.0 to 159.0] | 68.0 [32.0 to 137.0]
  Anti-HPV-18, CD4-d-TNFα, S+, Month 7: number analyzed (Participants) | 11 | 11
  Anti-HPV-18, CD4-d-TNFα, S+, Month 7 | 1337.0 [437.0 to 3141.0] | 1137.0 [648.0 to 2211.0]
  Anti-HPV-18, CD4-d-TNFα, S+, Month 12: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD4-d-TNFα, S+, Month 12 | 604.0 [391.0 to 1696.0] | 684.0 [443.0 to 1284.0]
  Anti-HPV-18, CD4-d-TNFα, S+, Month 24: number analyzed (Participants) | 10 | 12
  Anti-HPV-18, CD4-d-TNFα, S+, Month 24 | 601.0 [462.0 to 2122.0] | 768.5 [370.5 to 1673.0]
  Anti-HPV-18, CD4-d-TNFα, S+, Month 36: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD4-d-TNFα, S+, Month 36 | 652.5 [489.0 to 1590.0] | 444.0 [294.0 to 996.0]
  Anti-HPV-18, CD8-all doubles, S-, Day 0: number analyzed (Participants) | 77 | 69
  Anti-HPV-18, CD8-all doubles, S-, Day 0 | 11.0 [11.0 to 36.0] | 11.0 [11.0 to 33.0]
  Anti-HPV-18, CD8-all doubles, S-, Month 7: number analyzed (Participants) | 65 | 53
  Anti-HPV-18, CD8-all doubles, S-, Month 7 | 11.0 [11.0 to 37.0] | 11.0 [11.0 to 32.0]
  Anti-HPV-18, CD8 all doubles, S-, Month 12 | 28.0 [11.0 to 47.0] | 37.0 [11.0 to 51.5]
  Anti-HPV-18, CD8-all doubles, S-, Month 24: number analyzed (Participants) | 76 | 68
  Anti-HPV-18, CD8-all doubles, S-, Month 24 | 11.0 [11.0 to 51.0] | 11.0 [11.0 to 43.0]
  Anti-HPV-18, CD8-all doubles, S-, Month 36: number analyzed (Participants) | 72 | 56
  Anti-HPV-18, CD8-all doubles, S-, Month 36 | 32.0 [11.0 to 45.5] | 29.0 [11.0 to 51.0]
  Anti-HPV-18, CD8-all doubles, S+, Day 0: number analyzed (Participants) | 11 | 14
  Anti-HPV-18, CD8-all doubles, S+, Day 0 | 11.0 [11.0 to 27.0] | 11.0 [11.0 to 34.0]
  Anti-HPV-18, CD8-all doubles, S+, Month 7: number analyzed (Participants) | 11 | 11
  Anti-HPV-18, CD8-all doubles, S+, Month 7 | 11.0 [11.0 to 78.0] | 11.0 [11.0 to 73.0]
  Anti-HPV-18, CD8 all doubles, S+, Month 12: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD8 all doubles, S+, Month 12 | 44.0 [11.0 to 73.0] | 11.0 [11.0 to 33.0]
  Anti-HPV-18, CD8-all doubles, S+, Month 24: number analyzed (Participants) | 10 | 12
  Anti-HPV-18, CD8-all doubles, S+, Month 24 | 19.5 [11.0 to 47.0] | 11.0 [11.0 to 36.0]
  Anti-HPV-18, CD8-all doubles, S+, Month 36: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD8-all doubles, S+, Month 36 | 45.0 [11.0 to 85.0] | 34.0 [11.0 to 50.0]
  Anti-HPV-18, CD8-d-CD40L, S-, Day 0: number analyzed (Participants) | 77 | 69
  Anti-HPV-18, CD8-d-CD40L, S-, Day 0 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-CD40L, S-, Month 7: number analyzed (Participants) | 65 | 53
  Anti-HPV-18, CD8-d-CD40L, S-, Month 7 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-CD40L, S-, Month 12 | 7.0 [7.0 to 32.0] | 7.0 [7.0 to 36.5]
  Anti-HPV-18, CD8-d-CD40L, S-, Month 24: number analyzed (Participants) | 76 | 68
  Anti-HPV-18, CD8-d-CD40L, S-, Month 24 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-CD40L, S-, Month 36: number analyzed (Participants) | 72 | 56
  Anti-HPV-18, CD8-d-CD40L, S-, Month 36 | 7.0 [7.0 to 35.5] | 7.0 [7.0 to 37.5]
  Anti-HPV-18, CD8-d-CD40L, S+, Day 0: number analyzed (Participants) | 11 | 14
  Anti-HPV-18, CD8-d-CD40L, S+, Day 0 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-CD40L, S+, Month 7: number analyzed (Participants) | 11 | 11
  Anti-HPV-18, CD8-d-CD40L, S+, Month 7 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 27.0]
  Anti-HPV-18, CD8-d-CD40L, S+, Month 12: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD8-d-CD40L, S+, Month 12 | 34.5 [7.0 to 48.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-CD40L, S+, Month 24: number analyzed (Participants) | 10 | 12
  Anti-HPV-18, CD8-d-CD40L, S+, Month 24 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-CD40L, S+, Month 36: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD8-d-CD40L, S+, Month 36 | 25.0 [7.0 to 61.0] | 7.0 [7.0 to 30.0]
  Anti-HPV-18, CD8-d-IFNγ, S-, Day 0: number analyzed (Participants) | 77 | 69
  Anti-HPV-18, CD8-d-IFNγ, S-, Day 0 | 7.0 [7.0 to 29.0] | 7.0 [7.0 to 24.0]
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 7: number analyzed (Participants) | 65 | 53
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 7 | 7.0 [7.0 to 26.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 12 | 7.0 [7.0 to 34.0] | 7.0 [7.0 to 39.5]
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 24: number analyzed (Participants) | 76 | 68
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 24 | 7.0 [7.0 to 29.5] | 7.0 [7.0 to 33.5]
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 36: number analyzed (Participants) | 72 | 56
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 36 | 7.0 [7.0 to 40.5] | 7.0 [7.0 to 34.5]
  Anti-HPV-18, CD8-d-IFNγ, S+, Day 0: number analyzed (Participants) | 11 | 14
  Anti-HPV-18, CD8-d-IFNγ, S+, Day 0 | 7.0 [7.0 to 23.0] | 7.0 [7.0 to 30.0]
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 7: number analyzed (Participants) | 11 | 11
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 7 | 7.0 [7.0 to 74.0] | 7.0 [7.0 to 39.0]
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 12: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 12 | 16.0 [7.0 to 38.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 24: number analyzed (Participants) | 10 | 12
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 24 | 7.0 [7.0 to 9.0] | 7.0 [7.0 to 32.0]
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 36: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 36 | 7.0 [7.0 to 39.0] | 7.0 [7.0 to 40.0]
  Anti-HPV-18, CD8-d-IL-2, S-, Day 0: number analyzed (Participants) | 77 | 69
  Anti-HPV-18, CD8-d-IL-2, S-, Day 0 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IL-2, S-, Month 7: number analyzed (Participants) | 65 | 53
  Anti-HPV-18, CD8-d-IL-2, S-, Month 7 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IL-2, S-, Month 12 | 7.0 [7.0 to 26.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IL-2, S-, Month 24: number analyzed (Participants) | 76 | 68
  Anti-HPV-18, CD8-d-IL-2, S-, Month 24 | 7.0 [7.0 to 27.0] | 7.0 [7.0 to 14.5]
  Anti-HPV-18, CD8-d-IL-2, S-, Month 36: number analyzed (Participants) | 72 | 56
  Anti-HPV-18, CD8-d-IL-2, S-, Month 36 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IL-2, S+, Day 0: number analyzed (Participants) | 11 | 14
  Anti-HPV-18, CD8-d-IL-2, S+, Day 0 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IL-2, S+, Month 7: number analyzed (Participants) | 11 | 11
  Anti-HPV-18, CD8-d-IL-2, S+, Month 7 | 7.0 [7.0 to 24.0] | 7.0 [7.0 to 34.0]
  Anti-HPV-18, CD8-d-IL-2, S+, Month 12: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD8-d-IL-2, S+, Month 12 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 23.0]
  Anti-HPV-18, CD8-d-IL-2, S+, Month 24: number analyzed (Participants) | 10 | 12
  Anti-HPV-18, CD8-d-IL-2, S+, Month 24 | 7.0 [7.0 to 24.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IL-2, S+, Month 36: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD8-d-IL-2, S+, Month 36 | 7.0 [7.0 to 39.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-TNFα, S-, Day 0: number analyzed (Participants) | 77 | 69
  Anti-HPV-18, CD8-d-TNFα, S-, Day 0 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 8.0]
  Anti-HPV-18, CD8-d-TNFα, S-, Month 7: number analyzed (Participants) | 65 | 53
  Anti-HPV-18, CD8-d-TNFα, S-, Month 7 | 7.0 [7.0 to 31.0] | 7.0 [7.0 to 27.0]
  Anti-HPV-18, CD8-d-TNFα, S-, Month 12 | 7.0 [7.0 to 31.0] | 7.0 [7.0 to 35.0]
  Anti-HPV-18, CD8-d-TNFα, S-, Month 24: number analyzed (Participants) | 76 | 68
  Anti-HPV-18, CD8-d-TNFα, S-, Month 24 | 7.0 [7.0 to 32.5] | 7.0 [7.0 to 33.0]
  Anti-HPV-18, CD8-d-TNFα, S-, Month 36: number analyzed (Participants) | 72 | 56
  Anti-HPV-18, CD8-d-TNFα, S-, Month 36 | 7.0 [7.0 to 32.0] | 7.0 [7.0 to 35.0]
  Anti-HPV-18, CD8-d-TNFα, S+, Day 0: number analyzed (Participants) | 11 | 14
  Anti-HPV-18, CD8-d-TNFα, S+, Day 0 | 7.0 [7.0 to 23.0] | 7.0 [7.0 to 30.0]
  Anti-HPV-18, CD8-d-TNFα, S+, Month 7: number analyzed (Participants) | 11 | 11
  Anti-HPV-18, CD8-d-TNFα, S+, Month 7 | 7.0 [7.0 to 74.0] | 7.0 [7.0 to 62.0]
  Anti-HPV-18, CD8-d-TNFα, S+, Month 12: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD8-d-TNFα, S+, Month 12 | 7.0 [7.0 to 38.0] | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-TNFα, S+, Month 24: number analyzed (Participants) | 10 | 12
  Anti-HPV-18, CD8-d-TNFα, S+, Month 24 | 7.0 [7.0 to 31.0] | 7.0 [7.0 to 16.5]
  Anti-HPV-18, CD8-d-TNFα, S+, Month 36: number analyzed (Participants) | 10 | 13
  Anti-HPV-18, CD8-d-TNFα, S+, Month 36 | 17.0 [7.0 to 57.0] | 7.0 [7.0 to 29.0]

11. Secondary Outcome: Cell-mediated Immunogenicity Related to Anti-HPV-16 Specific T CMI Response for Cervarix 3 Group in a Sub-cohort of Subjects
Description: The CMI response represents the measure of the cytokines production (IL-2, IFN-γ, TNF-α, and CD40L) by HPV-antigen specific T lymphocytes and measured by ICS assay for HPV-16. The frequency was presented as a number of cytokine-positive cluster of differentiation (CD)4 i.e.CD4+/CD8+ cells per million CD4+/CD8+ cells. All doubles= T cell expressing at least 2 cytokines. Results were tabulated by the pre-vaccination status of the subjects, where S- = seronegative subjects (antibody concentration < cut-off value) prior to vaccination. S+ = seropositive subjects (antibody concentration ≥ cut-off value) prior to vaccination. The assay was performed on a subset of 100 subjects from Cervarix 3 Group.
Time Frame: At Day 0 and at Months 13, 18 and 36
Population: The analysis was based on the Month 36 ATP cohort for immunogenicity which included a sub-cohort of 100 subjects from Cervarix 3 Group, who returned for blood sampling at Month 36 and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination at the specified time points.
Measure: Median (Inter-Quartile Range); unit: cells/million T cells
Arm/Group | Cervarix 3 Group
Number analyzed (Participants) | 77
cells/million T cells
  Anti-HPV-16, CD4 all doubles, S-, Day 0 | 96.0 [61.0 to 170.0]
  Anti-HPV-16, CD4 all doubles, S-, Month 13: number analyzed (Participants) | 73
  Anti-HPV-16, CD4 all doubles, S-, Month 13 | 2399.0 [1514.0 to 4223.0]
  Anti-HPV-16, CD4 all doubles, S-, Month 18: number analyzed (Participants) | 73
  Anti-HPV-16, CD4 all doubles, S-, Month 18 | 1879.0 [1124.0 to 3449.0]
  Anti-HPV-16, CD4 all doubles, S-, Month 36: number analyzed (Participants) | 70
  Anti-HPV-16, CD4 all doubles, S-, Month 36 | 1786.5 [1064.0 to 3285.0]
  Anti-HPV-16, CD4 all doubles, S+, Day 0: number analyzed (Participants) | 7
  Anti-HPV-16, CD4 all doubles, S+, Day 0 | 169.0 [77.0 to 277.0]
  Anti-HPV-16, CD4 all doubles, S+, Month 13: number analyzed (Participants) | 6
  Anti-HPV-16, CD4 all doubles, S+, Month 13 | 2507.5 [1067.0 to 4212.0]
  Anti-HPV-16, CD4 all doubles, S+, Month 18: number analyzed (Participants) | 6
  Anti-HPV-16, CD4 all doubles, S+, Month 18 | 2717.5 [1597.0 to 4103.0]
  Anti-HPV-16, CD4 all doubles, S+, Month 36: number analyzed (Participants) | 7
  Anti-HPV-16, CD4 all doubles, S+, Month 36 | 1521.0 [297.0 to 3794.0]
  Anti-HPV-16, CD4-d-CD40L, S-, Day 0 | 89.0 [48.0 to 133.0]
  Anti-HPV-16, CD4-d-CD40L, S-, Month 13: number analyzed (Participants) | 73
  Anti-HPV-16, CD4-d-CD40L, S-, Month 13 | 2356.0 [1510.0 to 4165.0]
  Anti-HPV-16, CD4-d-CD40L, S-, Month 18: number analyzed (Participants) | 73
  Anti-HPV-16, CD4-d-CD40L, S-, Month 18 | 1831.0 [1070.0 to 3272.0]
  Anti-HPV-16, CD4-d-CD40L, S-, Month 36: number analyzed (Participants) | 70
  Anti-HPV-16, CD4-d-CD40L, S-, Month 36 | 1763.0 [1048.0 to 3239.0]
  Anti-HPV-16, CD4-d-CD40L, S+, Day 0: number analyzed (Participants) | 7
  Anti-HPV-16, CD4-d-CD40L, S+, Day 0 | 141.0 [73.0 to 261.0]
  Anti-HPV-16, CD4-d-CD40L, S+, Month 13: number analyzed (Participants) | 6
  Anti-HPV-16, CD4-d-CD40L, S+, Month 13 | 2450.5 [1036.0 to 4139.0]
  Anti-HPV-16, CD4-d-CD40L, S+, Month 18: number analyzed (Participants) | 6
  Anti-HPV-16, CD4-d-CD40L, S+, Month 18 | 2614.5 [1580.0 to 3862.0]
  Anti-HPV-16, CD4-d-CD40L, S+, Month 36: number analyzed (Participants) | 7
  Anti-HPV-16, CD4-d-CD40L, S+, Month 36 | 1426.0 [280.0 to 3697.0]
  Anti-HPV-16, CD4-d-IFNγ, S-, Day 0 | 35.0 [20.0 to 60.0]
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 13: number analyzed (Participants) | 73
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 13 | 651.0 [328.0 to 1356.0]
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 18: number analyzed (Participants) | 73
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 18 | 405.0 [208.0 to 821.0]
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 36: number analyzed (Participants) | 70
  Anti-HPV-16, CD4-d-IFNγ, S-, Month 36 | 646.0 [276.0 to 1282.0]
  Anti-HPV-16, CD4-d-IFNγ, S+, Day 0: number analyzed (Participants) | 7
  Anti-HPV-16, CD4-d-IFNγ, S+, Day 0 | 68.0 [33.0 to 203.0]
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 13: number analyzed (Participants) | 6
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 13 | 644.0 [204.0 to 1163.0]
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 18: number analyzed (Participants) | 6
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 18 | 708.5 [361.0 to 1218.0]
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 36: number analyzed (Participants) | 7
  Anti-HPV-16, CD4-d-IFNγ, S+, Month 36 | 310.0 [72.0 to 1783.0]
  Anti-HPV-16, CD4-d-IL-2, S-, Day 0 | 63.0 [34.0 to 111.0]
  Anti-HPV-16, CD4-d-IL-2, S-, Month 13: number analyzed (Participants) | 73
  Anti-HPV-16, CD4-d-IL-2, S-, Month 13 | 2220.0 [1406.0 to 4107.0]
  Anti-HPV-16, CD4-d-IL-2, S-, Month 18: number analyzed (Participants) | 73
  Anti-HPV-16, CD4-d-IL-2, S-, Month 18 | 1830.0 [1084.0 to 3221.0]
  Anti-HPV-16, CD4-d-IL-2, S-, Month 36: number analyzed (Participants) | 70
  Anti-HPV-16, CD4-d-IL-2, S-, Month 36 | 1670.5 [1009.0 to 3169.0]
  Anti-HPV-16, CD4-d-IL-2, S+, Day 0: number analyzed (Participants) | 7
  Anti-HPV-16, CD4-d-IL-2, S+, Day 0 | 121.0 [47.0 to 191.0]
  Anti-HPV-16, CD4-d-IL-2, S+, Month 13: number analyzed (Participants) | 6
  Anti-HPV-16, CD4-d-IL-2, S+, Month 13 | 2442.0 [835.0 to 4006.0]
  Anti-HPV-16, CD4-d-IL-2, S+, Month 18: number analyzed (Participants) | 6
  Anti-HPV-16, CD4-d-IL-2, S+, Month 18 | 2659.5 [1510.0 to 3870.0]
  Anti-HPV-16, CD4-d-IL-2, S+, Month 36: number analyzed (Participants) | 7
  Anti-HPV-16, CD4-d-IL-2, S+, Month 36 | 1028.0 [267.0 to 3629.0]
  Anti-HPV-16, CD4-d-TNFα, S-, Day 0 | 63.0 [37.0 to 99.0]
  Anti-HPV-16, CD4-d-TNFα, S-, Month 13: number analyzed (Participants) | 73
  Anti-HPV-16, CD4-d-TNFα, S-, Month 13 | 1643.0 [907.0 to 2988.0]
  Anti-HPV-16, CD4-d-TNFα, S-, Month 18: number analyzed (Participants) | 73
  Anti-HPV-16, CD4-d-TNFα, S-, Month 18 | 1326.0 [807.0 to 2627.0]
  Anti-HPV-16, CD4-d-TNFα, S-, Month 36: number analyzed (Participants) | 70
  Anti-HPV-16, CD4-d-TNFα, S-, Month 36 | 1300.5 [693.0 to 2267.0]
  Anti-HPV-16, CD4-d-TNFα, S+, Day 0: number analyzed (Participants) | 7
  Anti-HPV-16, CD4-d-TNFα, S+, Day 0 | 140.0 [32.0 to 164.0]
  Anti-HPV-16, CD4-d-TNFα, S+, Month 13: number analyzed (Participants) | 6
  Anti-HPV-16, CD4-d-TNFα, S+, Month 13 | 1843.0 [584.0 to 2657.0]
  Anti-HPV-16, CD4-d-TNFα, S+, Month 18: number analyzed (Participants) | 6
  Anti-HPV-16, CD4-d-TNFα, S+, Month 18 | 2085.0 [1380.0 to 2700.0]
  Anti-HPV-16, CD4-d-TNFα, S+, Month 36: number analyzed (Participants) | 7
  Anti-HPV-16, CD4-d-TNFα, S+, Month 36 | 1202.0 [169.0 to 2745.0]
  Anti-HPV-16, CD8-all doubles, S-, Day 0 | 27.0 [11.0 to 54.0]
  Anti-HPV-16, CD8-all doubles, S-, Month 13: number analyzed (Participants) | 73
  Anti-HPV-16, CD8-all doubles, S-, Month 13 | 11.0 [11.0 to 43.0]
  Anti-HPV-16, CD8-all doubles, S-, Month 18: number analyzed (Participants) | 73
  Anti-HPV-16, CD8-all doubles, S-, Month 18 | 11.0 [11.0 to 53.0]
  Anti-HPV-16, CD8-all doubles, S-, Month 36: number analyzed (Participants) | 70
  Anti-HPV-16, CD8-all doubles, S-, Month 36 | 21.5 [11.0 to 52.0]
  Anti-HPV-16, CD8-all doubles, S+, Day 0: number analyzed (Participants) | 7
  Anti-HPV-16, CD8-all doubles, S+, Day 0 | 33.0 [11.0 to 59.0]
  Anti-HPV-16, CD8-all doubles, S+, Month 13: number analyzed (Participants) | 6
  Anti-HPV-16, CD8-all doubles, S+, Month 13 | 43.0 [11.0 to 57.0]
  Anti-HPV-16, CD8-all doubles, S+, Month 18: number analyzed (Participants) | 6
  Anti-HPV-16, CD8-all doubles, S+, Month 18 | 27.0 [11.0 to 52.0]
  Anti-HPV-16, CD8-all doubles, S+, Month 36: number analyzed (Participants) | 7
  Anti-HPV-16, CD8-all doubles, S+, Month 36 | 11.0 [11.0 to 89.0]
  Anti-HPV-16, CD8-d-CD40L, S-, Day 0 | 7.0 [7.0 to 35.0]
  Anti-HPV-16, CD8-d-CD40L, S-, Month 13: number analyzed (Participants) | 73
  Anti-HPV-16, CD8-d-CD40L, S-, Month 13 | 7.0 [7.0 to 29.0]
  Anti-HPV-16, CD8-d-CD40L, S-, Month 18: number analyzed (Participants) | 73
  Anti-HPV-16, CD8-d-CD40L, S-, Month 18 | 7.0 [7.0 to 34.0]
  Anti-HPV-16, CD8-d-CD40L, S-, Month 36: number analyzed (Participants) | 70
  Anti-HPV-16, CD8-d-CD40L, S-, Month 36 | 7.0 [7.0 to 30.0]
  Anti-HPV-16, CD8-d-CD40L, S+, Day 0: number analyzed (Participants) | 7
  Anti-HPV-16, CD8-d-CD40L, S+, Day 0 | 7.0 [7.0 to 35.0]
  Anti-HPV-16, CD8-d-CD40L, S+, Month 13: number analyzed (Participants) | 6
  Anti-HPV-16, CD8-d-CD40L, S+, Month 13 | 7.0 [7.0 to 34.0]
  Anti-HPV-16, CD8-d-CD40L, S+, Month 18: number analyzed (Participants) | 6
  Anti-HPV-16, CD8-d-CD40L, S+, Month 18 | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-CD40L, S+, Month 36: number analyzed (Participants) | 7
  Anti-HPV-16, CD8-d-CD40L, S+, Month 36 | 7.0 [7.0 to 46.0]
  Anti-HPV-16, CD8-d-IFNγ, S-, Day 0 | 7.0 [7.0 to 44.0]
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 13: number analyzed (Participants) | 73
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 13 | 7.0 [7.0 to 35.0]
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 18: number analyzed (Participants) | 73
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 18 | 7.0 [7.0 to 37.0]
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 36: number analyzed (Participants) | 70
  Anti-HPV-16, CD8-d-IFNγ, S-, Month 36 | 7.0 [7.0 to 38.0]
  Anti-HPV-16, CD8-d-IFNγ, S+, Day 0: number analyzed (Participants) | 7
  Anti-HPV-16, CD8-d-IFNγ, S+, Day 0 | 29.0 [7.0 to 55.0]
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 13: number analyzed (Participants) | 6
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 13 | 25.5 [7.0 to 53.0]
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 18: number analyzed (Participants) | 6
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 18 | 7.0 [7.0 to 33.0]
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 36: number analyzed (Participants) | 7
  Anti-HPV-16, CD8-d-IFNγ, S+, Month 36 | 7.0 [7.0 to 46.0]
  Anti-HPV-16, CD8-d-IL-2, S-, Day 0 | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-IL-2, S-, Month 13: number analyzed (Participants) | 73
  Anti-HPV-16, CD8-d-IL-2, S-, Month 13 | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-IL-2, S-, Month 18: number analyzed (Participants) | 73
  Anti-HPV-16, CD8-d-IL-2, S-, Month 18 | 7.0 [7.0 to 29.0]
  Anti-HPV-16, CD8-d-IL-2, S-, Month 36: number analyzed (Participants) | 70
  Anti-HPV-16, CD8-d-IL-2, S-, Month 36 | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-IL-2, S+, Day 0: number analyzed (Participants) | 7
  Anti-HPV-16, CD8-d-IL-2, S+, Day 0 | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-IL-2, S+, Month 13: number analyzed (Participants) | 6
  Anti-HPV-16, CD8-d-IL-2, S+, Month 13 | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-IL-2, S+, Month 18: number analyzed (Participants) | 6
  Anti-HPV-16, CD8-d-IL-2, S+, Month 18 | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-IL-2, S+, Month 36: number analyzed (Participants) | 7
  Anti-HPV-16, CD8-d-IL-2, S+, Month 36 | 7.0 [7.0 to 46.0]
  Anti-HPV-16, CD8-d-TNFα, S-, Day 0 | 7.0 [7.0 to 27.0]
  Anti-HPV-16, CD8-d-TNFα, S-, Month 13: number analyzed (Participants) | 73
  Anti-HPV-16, CD8-d-TNFα, S-, Month 13 | 7.0 [7.0 to 29.0]
  Anti-HPV-16, CD8-d-TNFα, S-, Month 18: number analyzed (Participants) | 73
  Anti-HPV-16, CD8-d-TNFα, S-, Month 18 | 7.0 [7.0 to 41.0]
  Anti-HPV-16, CD8-d-TNFα, S-, Month 36: number analyzed (Participants) | 70
  Anti-HPV-16, CD8-d-TNFα, S-, Month 36 | 7.0 [7.0 to 38.0]
  Anti-HPV-16, CD8-d-TNFα, S+, Day 0: number analyzed (Participants) | 7
  Anti-HPV-16, CD8-d-TNFα, S+, Day 0 | 7.0 [7.0 to 7.0]
  Anti-HPV-16, CD8-d-TNFα, S+, Month 13: number analyzed (Participants) | 6
  Anti-HPV-16, CD8-d-TNFα, S+, Month 13 | 20.5 [7.0 to 44.0]
  Anti-HPV-16, CD8-d-TNFα, S+, Month 18: number analyzed (Participants) | 6
  Anti-HPV-16, CD8-d-TNFα, S+, Month 18 | 20.0 [7.0 to 39.0]
  Anti-HPV-16, CD8-d-TNFα, S+, Month 36: number analyzed (Participants) | 7
  Anti-HPV-16, CD8-d-TNFα, S+, Month 36 | 7.0 [7.0 to 7.0]

12. Secondary Outcome: Cell-mediated Immunogenicity Related to Anti-HPV-18 Specific T CMI Response for Cervarix 3 Group in a Sub-cohort of Subjects
Description: The CMI response represents the measure of the cytokines production (i.e. IL-2, IFN-γ, TNF-α, and CD40L) by HPV-antigen specific T lymphocytes and measured by ICS assay for HPV-18. The frequency was presented as a number of cytokine-producing CD4+/CD8+ cells per million CD4+/CD8+ cells. All doubles = T cell expressing at least 2 cytokines. Results were tabulated by the pre-vaccination status of the subjects, where S- = seronegative subjects (antibody concentration < cut-off value) prior to vaccination. S+ = seropositive subjects (antibody concentration ≥ cut-off value) prior to vaccination. The assay was performed on a subset of 100 subjects from Cervarix 3 Group.
Time Frame: At Day 0 and at Months 13, 18 and 36
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: cells/million T-cells
Arm/Group | Cervarix 3 Group
Number analyzed (Participants) | 82
cells/million T-cells
  Anti-HPV-18, CD4 all doubles, S-, Day 0 | 99.0 [61.0 to 149.0]
  Anti-HPV-18, CD4 all doubles, S-, Month 13: number analyzed (Participants) | 77
  Anti-HPV-18, CD4 all doubles, S-, Month 13 | 1499.0 [1033.0 to 2928.0]
  Anti-HPV-18, CD4 all doubles, S-, Month 18: number analyzed (Participants) | 77
  Anti-HPV-18, CD4 all doubles, S-, Month 18 | 1222.0 [796.0 to 2116.0]
  Anti-HPV-18, CD4 all doubles, S-, Month 36: number analyzed (Participants) | 75
  Anti-HPV-18, CD4 all doubles, S-, Month 36 | 1158.0 [606.0 to 2185.0]
  Anti-HPV-18, CD4 all doubles, S+, Day 0: number analyzed (Participants) | 2
  Anti-HPV-18, CD4 all doubles, S+, Day 0 | 107.5 [69.0 to 146.0]
  Anti-HPV-18, CD4 all doubles, S+, Month 13: number analyzed (Participants) | 2
  Anti-HPV-18, CD4 all doubles, S+, Month 13 | 1968.5 [1753.0 to 2184.0]
  Anti-HPV-18, CD4 all doubles, S+, Month 18: number analyzed (Participants) | 2
  Anti-HPV-18, CD4 all doubles, S+, Month 18 | 1250.0 [1156.0 to 1344.0]
  Anti-HPV-18, CD4 all doubles, S+, Month 36: number analyzed (Participants) | 2
  Anti-HPV-18, CD4 all doubles, S+, Month 36 | 1399.5 [1004.0 to 1795.0]
  Anti-HPV-18, CD4-d-CD40L, S-, Day 0 | 82.5 [42.0 to 125.0]
  Anti-HPV-18, CD4-d-CD40L, S-, Month 13: number analyzed (Participants) | 77
  Anti-HPV-18, CD4-d-CD40L, S-, Month 13 | 1472.0 [1003.0 to 2880.0]
  Anti-HPV-18, CD4-d-CD40L, S-, Month 18: number analyzed (Participants) | 77
  Anti-HPV-18, CD4-d-CD40L, S-, Month 18 | 1199.0 [748.0 to 2098.0]
  Anti-HPV-18, CD4-d-CD40L, S-, Month 36: number analyzed (Participants) | 75
  Anti-HPV-18, CD4-d-CD40L, S-, Month 36 | 1154.0 [563.0 to 2157.0]
  Anti-HPV-18, CD4-d-CD40L, S+, Day 0: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-CD40L, S+, Day 0 | 103.5 [65.0 to 142.0]
  Anti-HPV-18, CD4-d-CD40L, S+, Month 13: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-CD40L, S+, Month 13 | 1904.5 [1656.0 to 2153.0]
  Anti-HPV-18, CD4-d-CD40L, S+, Month 18: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-CD40L, S+, Month 18 | 1174.5 [1110.0 to 1239.0]
  Anti-HPV-18, CD4-d-CD40L, S+, Month 36: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-CD40L, S+, Month 36 | 1320.0 [918.0 to 1722.0]
  Anti-HPV-18, CD4-d-IFNγ, S-, Day 0 | 35.0 [23.0 to 61.0]
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 13: number analyzed (Participants) | 77
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 13 | 349.0 [173.0 to 1221.0]
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 18: number analyzed (Participants) | 77
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 18 | 226.0 [108.0 to 575.0]
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 36: number analyzed (Participants) | 75
  Anti-HPV-18, CD4-d-IFNγ, S-, Month 36 | 318.0 [140.0 to 766.0]
  Anti-HPV-18, CD4-d-IFNγ, S+, Day 0: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-IFNγ, S+, Day 0 | 33.5 [24.0 to 43.0]
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 13: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 13 | 378.0 [307.0 to 449.0]
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 18: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 18 | 157.5 [136.0 to 179.0]
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 36: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-IFNγ, S+, Month 36 | 389.0 [231.0 to 547.0]
  Anti-HPV-18, CD4-d-IL-2, S-, Day 0 | 58.5 [32.0 to 98.0]
  Anti-HPV-18, CD4-d-IL-2, S-, Month 13: number analyzed (Participants) | 77
  Anti-HPV-18, CD4-d-IL-2, S-, Month 13 | 1398.0 [812.0 to 2743.0]
  Anti-HPV-18, CD4-d-IL-2, S-, Month 18: number analyzed (Participants) | 77
  Anti-HPV-18, CD4-d-IL-2, S-, Month 18 | 1102.0 [719.0 to 1924.0]
  Anti-HPV-18, CD4-d-IL-2, S-, Month 36: number analyzed (Participants) | 75
  Anti-HPV-18, CD4-d-IL-2, S-, Month 36 | 1086.0 [535.0 to 1974.0]
  Anti-HPV-18, CD4-d-IL-2, S+, Day 0: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-IL-2, S+, Day 0 | 46.5 [33.0 to 60.0]
  Anti-HPV-18, CD4-d-IL-2, S+, Month 13: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-IL-2, S+, Month 13 | 1845.0 [1544.0 to 2146.0]
  Anti-HPV-18, CD4-d-IL-2, S+, Month 18: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-IL-2, S+, Month 18 | 1151.0 [1078.0 to 1224.0]
  Anti-HPV-18, CD4-d-IL-2, S+, Month 36: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-IL-2, S+, Month 36 | 1160.0 [827.0 to 1493.0]
  Anti-HPV-18, CD4-d-TNFα, S-, Day 0 | 60.5 [34.0 to 97.0]
  Anti-HPV-18, CD4-d-TNFα, S-, Month 13: number analyzed (Participants) | 77
  Anti-HPV-18, CD4-d-TNFα, S-, Month 13 | 1029.0 [649.0 to 2051.0]
  Anti-HPV-18, CD4-d-TNFα, S-, Month 18: number analyzed (Participants) | 77
  Anti-HPV-18, CD4-d-TNFα, S-, Month 18 | 921.0 [539.0 to 1783.0]
  Anti-HPV-18, CD4-d-TNFα, S-, Month 36: number analyzed (Participants) | 75
  Anti-HPV-18, CD4-d-TNFα, S-, Month 36 | 812.0 [384.0 to 1545.0]
  Anti-HPV-18, CD4-d-TNFα, S+, Day 0: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-TNFα, S+, Day 0 | 66.5 [29.0 to 104.0]
  Anti-HPV-18, CD4-d-TNFα, S+, Month 13: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-TNFα, S+, Month 13 | 1449.5 [1317.0 to 1582.0]
  Anti-HPV-18, CD4-d-TNFα, S+, Month 18: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-TNFα, S+, Month 18 | 954.5 [873.0 to 1036.0]
  Anti-HPV-18, CD4-d-TNFα, S+, Month 36: number analyzed (Participants) | 2
  Anti-HPV-18, CD4-d-TNFα, S+, Month 36 | 1127.0 [847.0 to 1407.0]
  Anti-HPV-18, CD8-all doubles, S-, Day 0 | 11.0 [11.0 to 47.0]
  Anti-HPV-18, CD8-all doubles, S-, Month 13: number analyzed (Participants) | 77
  Anti-HPV-18, CD8-all doubles, S-, Month 13 | 32.0 [11.0 to 49.0]
  Anti-HPV-18, CD8-all doubles, S-, Month 18: number analyzed (Participants) | 77
  Anti-HPV-18, CD8-all doubles, S-, Month 18 | 34.0 [11.0 to 50.0]
  Anti-HPV-18, CD8-all doubles, S-, Month 36: number analyzed (Participants) | 75
  Anti-HPV-18, CD8-all doubles, S-, Month 36 | 33.0 [11.0 to 56.0]
  Anti-HPV-18, CD8-all doubles, S+, Day 0: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-all doubles, S+, Day 0 | 29.0 [11.0 to 47.0]
  Anti-HPV-18, CD8-all doubles, S+, Month 13: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-all doubles, S+, Month 13 | 63.5 [39.0 to 88.0]
  Anti-HPV-18, CD8-all doubles, S+, Month 18: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-all doubles, S+, Month 18 | 11.0 [11.0 to 11.0]
  Anti-HPV-18, CD8-all doubles, S+, Month 36: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-all doubles, S+, Month 36 | 45.0 [11.0 to 79.0]
  Anti-HPV-18, CD8-d-CD40L, S-, Day 0 | 7.0 [7.0 to 30.0]
  Anti-HPV-18, CD8-d-CD40L, S-, Month 13: number analyzed (Participants) | 77
  Anti-HPV-18, CD8-d-CD40L, S-, Month 13 | 7.0 [7.0 to 38.0]
  Anti-HPV-18, CD8-d-CD40L, S-, Month 18: number analyzed (Participants) | 77
  Anti-HPV-18, CD8-d-CD40L, S-, Month 18 | 7.0 [7.0 to 34.0]
  Anti-HPV-18, CD8-d-CD40L, S-, Month 36: number analyzed (Participants) | 75
  Anti-HPV-18, CD8-d-CD40L, S-, Month 36 | 7.0 [7.0 to 38.0]
  Anti-HPV-18, CD8-d-CD40L, S+, Day 0: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-CD40L, S+, Day 0 | 25.0 [7.0 to 43.0]
  Anti-HPV-18, CD8-d-CD40L, S+, Month 13: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-CD40L, S+, Month 13 | 21.0 [7.0 to 35.0]
  Anti-HPV-18, CD8-d-CD40L, S+, Month 18: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-CD40L, S+, Month 18 | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-CD40L, S+, Month 36: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-CD40L, S+, Month 36 | 41.0 [7.0 to 75.0]
  Anti-HPV-18, CD8-d-IFNγ, S-, Day 0 | 7.0 [7.0 to 41.0]
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 13: number analyzed (Participants) | 77
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 13 | 7.0 [7.0 to 40.0]
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 18: number analyzed (Participants) | 77
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 18 | 7.0 [7.0 to 37.0]
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 36: number analyzed (Participants) | 75
  Anti-HPV-18, CD8-d-IFNγ, S-, Month 36 | 7.0 [7.0 to 44.0]
  Anti-HPV-18, CD8-d-IFNγ, S+, Day 0: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-IFNγ, S+, Day 0 | 25.0 [7.0 to 43.0]
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 13: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 13 | 59.5 [35.0 to 84.0]
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 18: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 18 | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 36: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-IFNγ, S+, Month 36 | 41.0 [7.0 to 75.0]
  Anti-HPV-18, CD8-d-IL-2, S-, Day 0 | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IL-2, S-, Month 13: number analyzed (Participants) | 77
  Anti-HPV-18, CD8-d-IL-2, S-, Month 13 | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IL-2, S-, Month 18: number analyzed (Participants) | 77
  Anti-HPV-18, CD8-d-IL-2, S-, Month 18 | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IL-2, S-, Month 36: number analyzed (Participants) | 75
  Anti-HPV-18, CD8-d-IL-2, S-, Month 36 | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IL-2, S+, Day 0: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-IL-2, S+, Day 0 | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IL-2, S+, Month 13: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-IL-2, S+, Month 13 | 45.5 [7.0 to 84.0]
  Anti-HPV-18, CD8-d-IL-2, S+, Month 18: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-IL-2, S+, Month 18 | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-IL-2, S+, Month 36: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-IL-2, S+, Month 36 | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-TNFα, S-, Day 0 | 7.0 [7.0 to 38.0]
  Anti-HPV-18, CD8-d-TNFα, S-, Month 13: number analyzed (Participants) | 77
  Anti-HPV-18, CD8-d-TNFα, S-, Month 13 | 7.0 [7.0 to 30.0]
  Anti-HPV-18, CD8-d-TNFα, S-, Month 18: number analyzed (Participants) | 77
  Anti-HPV-18, CD8-d-TNFα, S-, Month 18 | 7.0 [7.0 to 40.0]
  Anti-HPV-18, CD8-d-TNFα, S-, Month 36: number analyzed (Participants) | 75
  Anti-HPV-18, CD8-d-TNFα, S-, Month 36 | 7.0 [7.0 to 35.0]
  Anti-HPV-18, CD8-d-TNFα, S+, Day 0: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-TNFα, S+, Day 0 | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-TNFα, S+, Month 13: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-TNFα, S+, Month 13 | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-TNFα, S+, Month 18: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-TNFα, S+, Month 18 | 7.0 [7.0 to 7.0]
  Anti-HPV-18, CD8-d-TNFα, S+, Month 36: number analyzed (Participants) | 2
  Anti-HPV-18, CD8-d-TNFα, S+, Month 36 | 7.0 [7.0 to 7.0]

13. Secondary Outcome: Cell-mediated Immunogenicity Related to Anti-HPV-16 Specific B CMI Response for Cervarix 1 Group and Cervarix 2 Group in a Sub-cohort of Subjects
Description: The CMI response was assessed as being the frequency of B-cell memory of HPV-16 antigen-specific memory B-cells per million memory B-cells in subjects with detectable B-cells. The results are presented by pre-vaccination status, where S- = seronegative subjects (antibody concentration < cut-off value) prior to vaccination and S+ = seropositive subjects (antibody concentration ≥ cut-off value) prior to vaccination. The assay was performed on a subset of 100 subjects per study group.
Time Frame: At Day 0 and at Months 7, 12, 24 and 36
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: cells/million B-cells
Arm/Group | Cervarix 1 Group | Cervarix 2 Group
Number analyzed (Participants) | 75 | 63
cells/million B-cells
  Anti-HPV-16, S-, Day 0: number analyzed (Participants) | 74 | 63
  Anti-HPV-16, S-, Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Anti-HPV-16, S-, Month 7: number analyzed (Participants) | 70 | 46
  Anti-HPV-16, S-, Month 7 | 2155.0 [886.0 to 5421.0] | 1510.0 [799.0 to 3114.0]
  Anti-HPV-16, S-, Month 12: number analyzed (Participants) | 55 | 42
  Anti-HPV-16, S-, Month 12 | 801.0 [361.0 to 2648.0] | 1145.0 [371.0 to 3215.0]
  Anti-HPV-16, S-, Month 24: number analyzed (Participants) | 75 | 60
  Anti-HPV-16, S-, Month 24 | 318.0 [95.0 to 697.0] | 594.5 [147.5 to 1133.5]
  Anti-HPV-16, S-, Month 36: number analyzed (Participants) | 70 | 53
  Anti-HPV-16, S-, Month 36 | 560.5 [157.0 to 1012.0] | 448.0 [219.0 to 821.0]
  Anti-HPV-16, S+, Day 0: number analyzed (Participants) | 8 | 13
  Anti-HPV-16, S+, Day 0 | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 51.0]
  Anti-HPV-16, S+, Month 7: number analyzed (Participants) | 7 | 11
  Anti-HPV-16, S+, Month 7 | 4838.0 [1513.0 to 11824.0] | 477.0 [139.0 to 4928.0]
  Anti-HPV-16, S+, Month 12: number analyzed (Participants) | 2 | 9
  Anti-HPV-16, S+, Month 12 | 5056.0 [5018.0 to 5094.0] | 539.0 [340.0 to 2111.0]
  Anti-HPV-16, S+, Month 24: number analyzed (Participants) | 8 | 12
  Anti-HPV-16, S+, Month 24 | 621.0 [324.5 to 1751.5] | 568.5 [50.0 to 1955.0]
  Anti-HPV-16, S+, Month 36: number analyzed (Participants) | 6 | 13
  Anti-HPV-16, S+, Month 36 | 475.0 [414.0 to 822.0] | 107.0 [1.0 to 1275.0]

14. Secondary Outcome: Cell-mediated Immunogenicity Related to Anti-HPV-18 Specific B CMI Response for Cervarix 1 Group and Cervarix 2 Group in a Sub-cohort of Subjects
Description: The cell-mediated immune response was assessed as being the frequency of B-cell memory of HPV-18 antigen-specific memory B-cells per million memory B-cells in subjects with detectable B-cells. The results are presented by pre-vaccination status, where S- = seronegative subjects (antibody concentration < cut-off value) prior to vaccination and S+ = seropositive subjects (antibody concentration ≥ cut-off value) prior to vaccination. The assay was performed on a subset of 100 subjects per study group.
Time Frame: At Day 0 and at Months 7, 12, 24 and 36
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: cells/million B-cells
Arm/Group | Cervarix 1 Group | Cervarix 2 Group
Number analyzed (Participants) | 72 | 63
cells/million B-cells
  Anti-HPV-18, S-, Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Anti-HPV-18, S-, Month 7: number analyzed (Participants) | 67 | 48
  Anti-HPV-18, S-, Month 7 | 958.0 [386.0 to 2500.0] | 817.5 [368.0 to 1894.5]
  Anti-HPV-18, S-, Month 24: number analyzed (Participants) | 72 | 61
  Anti-HPV-18, S-, Month 24 | 236.0 [61.5 to 710.0] | 274.0 [71.0 to 829.0]
  Anti-HPV-18, S-, Month 36: number analyzed (Participants) | 67 | 54
  Anti-HPV-18, S-, Month 36 | 269.0 [62.0 to 732.0] | 284.5 [90.0 to 582.0]
  Anti-HPV-18, S+, Day 0: number analyzed (Participants) | 10 | 14
  Anti-HPV-18, S+, Day 0 | 1.0 [1.0 to 44.0] | 1.0 [1.0 to 22.0]
  Anti-HPV-18, S+, Month 7: number analyzed (Participants) | 10 | 10
  Anti-HPV-18, S+, Month 7 | 2016.5 [423.0 to 2797.0] | 439.5 [31.0 to 1779.0]
  Anti-HPV-18, S+, Month 24: number analyzed (Participants) | 11 | 12
  Anti-HPV-18, S+, Month 24 | 299.0 [117.0 to 643.0] | 338.5 [174.0 to 786.0]
  Anti-HPV-18, S+, Month 36: number analyzed (Participants) | 9 | 12
  Anti-HPV-18, S+, Month 36 | 154.0 [141.0 to 427.0] | 93.0 [18.0 to 762.0]

15. Secondary Outcome: Cell-mediated Immunogenicity Related to Anti-HPV-16 Specific B CMI Response for Cervarix 3 Group in a Sub-cohort of Subjects
Description: The cell-mediated immune response was assessed as being the frequency of B-cell memory of HPV-16 antigen-specific memory B-cells per million memory B-cells in subjects with detectable B-cells. The results are presented by pre-vaccination status, where S- = seronegative subjects (antibody concentration < cut-off value) prior to vaccination and S+ = seropositive subjects (antibody concentration ≥ cut-off value) prior to vaccination. The assay was performed on a subset of 100 subjects from Cervarix 3 Group.
Time Frame: At Day 0 and at Months 13, 18 and 36
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: cells/million B-cells
Arm/Group | Cervarix 3 Group
Number analyzed (Participants) | 68
cells/million B-cells
  Anti-HPV-16, S-, Day 0: number analyzed (Participants) | 66
  Anti-HPV-16, S-, Day 0 | 1.0 [1.0 to 7.0]
  Anti-HPV-16, S-, Month 13 | 2809.5 [1402.5 to 5045.5]
  Anti-HPV-16, S-, Month 18: number analyzed (Participants) | 60
  Anti-HPV-16, S-, Month 18 | 766.0 [412.0 to 1946.5]
  Anti-HPV-16, S-, Month 36: number analyzed (Participants) | 67
  Anti-HPV-16, S-, Month 36 | 613.0 [322.0 to 1301.0]
  Anti-HPV-16, S+, Day 0: number analyzed (Participants) | 5
  Anti-HPV-16, S+, Day 0 | 1.0 [1.0 to 20.0]
  Anti-HPV-16, S+, Month 13: number analyzed (Participants) | 5
  Anti-HPV-16, S+, Month 13 | 5996.0 [919.0 to 7353.0]
  Anti-HPV-16, S+, Month 18: number analyzed (Participants) | 5
  Anti-HPV-16, S+, Month 18 | 2130.0 [808.0 to 2271.0]
  Anti-HPV-16, S+, Month 36: number analyzed (Participants) | 6
  Anti-HPV-16, S+, Month 36 | 425.0 [102.0 to 714.0]

16. Secondary Outcome: Cell-mediated Immunogenicity Related to Anti-HPV-18 Specific B CMI Response for Cervarix 3 Group in a Sub-cohort of Subjects
Description: The cell-mediated immune response was assessed as being the frequency of B-cell memory of HPV-18 antigen-specific memory B-cells per million memory B-cells in subjects with detectable B-cells. The results are presented by pre-vaccination status, where S- = seronegative subjects (antibody concentration < cut-off value) prior to vaccination and S+ = seropositive subjects (antibody concentration ≥ cut off value) prior to vaccination. The assay was performed on a subset of 100 subjects from Cervarix 3 Group.
Time Frame: At Day 0 and at Months 13, 18 and 36
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: cells/million B-cells
Arm/Group | Cervarix 3 Group
Number analyzed (Participants) | 72
cells/million B-cells
  Anti-HPV-18, S-, Day 0: number analyzed (Participants) | 70
  Anti-HPV-18, S-, Day 0 | 1.0 [1.0 to 1.0]
  Anti-HPV-18, S-, Month 13: number analyzed (Participants) | 71
  Anti-HPV-18, S-, Month 13 | 1165.0 [602.0 to 1660.0]
  Anti-HPV-18, S-, Month 18: number analyzed (Participants) | 64
  Anti-HPV-18, S-, Month 18 | 561.5 [132.0 to 1213.5]
  Anti-HPV-18, S-, Month 36 | 361.0 [112.0 to 724.0]
  Anti-HPV-18, S+, Day 0: number analyzed (Participants) | 1
  Anti-HPV-18, S+, Day 0 | 48.0 [48.0 to 48.0]
  Anti-HPV-18, S+, Month 13: number analyzed (Participants) | 2
  Anti-HPV-18, S+, Month 13 | 758.0 [114.0 to 1402.0]
  Anti-HPV-18, S+, Month 18: number analyzed (Participants) | 1
  Anti-HPV-18, S+, Month 18 | 938.0 [938.0 to 938.0]
  Anti-HPV-18, S+, Month 36: number analyzed (Participants) | 1
  Anti-HPV-18, S+, Month 36 | 1231.0 [1231.0 to 1231.0]

17. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any solicited local symptom regardless of their intensity grade. Grade 3 pain = significant pain at rest, that prevented normal every day activity. Grade 3 redness/swelling = redness/swelling above 50 millimeters (mm).
Time Frame: During the 7-day period (Days 0-6) after each vaccine dose and across doses
Population: The analysis was based on the Total Vaccinated Cohort (TVC), which included all vaccinated subjects who received at least one dose of vaccine and for whom data were available and symptom sheet completed. Subjects from Cervarix 1 and Cervarix 3 Groups received only 2 doses of vaccine, therefore data are presented up to Dose 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group
Number analyzed (Participants) | 550 | 480 | 413
Participants
  Any Pain - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Any Pain - Dose 1 | 461 | 439 | 354
  Grade 3 Pain - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Grade 3 Pain - Dose 1 | 24 | 21 | 21
  Any Pain - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Any Pain - Dose 2 | 446 | 377 | 323
  Grade 3 Pain - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Grade 3 Pain - Dose 2 | 33 | 25 | 31
  Any Pain - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Any Pain - Dose 3 |  | 358 |
  Grade 3 Pain - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Grade 3 Pain - Dose 3 |  | 20 |
  Any Pain - Across doses | 499 | 461 | 381
  Grade 3 Pain - Across doses | 50 | 53 | 48
  Any Redness - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Any Redness - Dose 1 | 167 | 135 | 126
  Grade 3 Redness - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Grade 3 Redness - Dose 1 | 0 | 2 | 2
  Any Redness - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Any Redness - Dose 2 | 180 | 143 | 153
  Grade 3 Redness - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Grade 3 Redness - Dose 2 | 4 | 5 | 1
  Any Redness - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Any Redness - Dose 3 |  | 142 |
  Grade 3 Redness - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Grade 3 Redness - Dose 3 |  | 5 |
  Any Redness - Across doses | 247 | 212 | 197
  Grade 3 Redness - Across doses | 4 | 10 | 3
  Any Swelling - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Any Swelling - Dose 1 | 141 | 105 | 101
  Grade 3 Swelling - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Grade 3 Swelling - Dose 1 | 3 | 1 | 4
  Any Swelling - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Any Swelling - Dose 2 | 166 | 131 | 135
  Grade 3 Swelling - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Grade 3 Swelling - Dose 2 | 2 | 4 | 2
  Any Swelling - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Any Swelling - Dose 3 |  | 136 |
  Grade 3 Swelling - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Grade 3 Swelling - Dose 3 |  | 3 |
  Any Swelling - Across doses | 225 | 204 | 171
  Grade 3 Swelling - Across doses | 5 | 6 | 6

18. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, rash, fever and urticaria. Any = occurrence of any solicited general symptom regardless of intensity grade or relationship to vaccination. Any fever = axillary temperature ≥ 37.5 degrees Celsius (°C). Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever greater than (>) 39.0 °C. Related = general symptom assessed by the investigator as causally related to the vaccination.
Time Frame: During the 7-day period (Days 0-6) after each vaccine dose and across doses
Population: The analysis was based on the TVC, which included all vaccinated subjects who received at least one dose of vaccine and for whom data were available and symptom sheet completed. Subjects from Cervarix 1 and Cervarix 3 Groups received only 2 doses of vaccine, therefore data are presented up to Dose 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group
Number analyzed (Participants) | 550 | 480 | 413
Participants
  Any Artharlgia - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Any Artharlgia - Dose 1 | 61 | 53 | 52
  Grade 3 Arthralgia - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Grade 3 Arthralgia - Dose 1 | 8 | 3 | 3
  Related Arthralgia - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Related Arthralgia - Dose 1 | 56 | 50 | 45
  Any Artharlgia - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Any Artharlgia - Dose 2 | 71 | 56 | 64
  Grade 3 Arthralgia - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Grade 3 Arthralgia - Dose 2 | 2 | 1 | 3
  Related Arthralgia - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Related Arthralgia - Dose 2 | 64 | 50 | 57
  Any Artharlgia - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Any Artharlgia - Dose 3 |  | 49 |
  Grade 3 Arthralgia - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Grade 3 Arthralgia - Dose 3 |  | 3 |
  Related Arthralgia - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Related Arthralgia - Dose 3 |  | 42 |
  Any Artharlgia - Across doses | 111 | 107 | 93
  Grade 3 Arthralgia - Across doses | 9 | 6 | 6
  Related Arthralgia - Across doses | 105 | 102 | 83
  Any Fatigue - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Any Fatigue - Dose 1 | 181 | 238 | 156
  Grade 3 Fatigue - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Grade 3 Fatigue - Dose 1 | 7 | 9 | 10
  Related Fatigue - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Related Fatigue - Dose 1 | 153 | 205 | 129
  Any Fatigue - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Any Fatigue - Dose 2 | 167 | 168 | 144
  Grade 3 Fatigue - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Grade 3 Fatigue - Dose 2 | 9 | 11 | 14
  Related Fatigue - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Related Fatigue - Dose 2 | 149 | 142 | 119
  Any Fatigue - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Any Fatigue - Dose 3 |  | 177 |
  Grade 3 Fatigue - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Grade 3 Fatigue - Dose 3 |  | 12 |
  Related Fatigue - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Related Fatigue - Dose 3 |  | 161 |
  Any Fatigue - Across doses | 247 | 310 | 215
  Grade 3 Fatigue - Across doses | 14 | 25 | 21
  Related Fatigue - Across doses | 221 | 294 | 185
  Any Gastrointestinal - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Any Gastrointestinal - Dose 1 | 59 | 88 | 44
  Grade 3 Gastrointestinal - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Grade 3 Gastrointestinal - Dose 1 | 1 | 2 | 3
  Related Gastrointestinal - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Related Gastrointestinal - Dose 1 | 49 | 67 | 32
  Any Gastrointestinal - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Any Gastrointestinal - Dose 2 | 51 | 50 | 48
  Grade 3 Gastrointestinal - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Grade 3 Gastrointestinal - Dose 2 | 6 | 2 | 4
  Related Gastrointestinal - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Related Gastrointestinal - Dose 2 | 34 | 36 | 40
  Any Gastrointestinal - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Any Gastrointestinal - Dose 3 |  | 45 |
  Grade 3 Gastrointestinal - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Grade 3 Gastrointestinal - Dose 3 |  | 7 |
  Related Gastrointestinal - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Related Gastrointestinal - Dose 3 |  | 35 |
  Any Gastrointestinal - Across doses | 98 | 134 | 77
  Grade 3 Gastrointestinal - Across doses | 7 | 11 | 7
  Related Gastrointestinal - Across doses | 77 | 106 | 62
  Any Headache - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Any Headache - Dose 1 | 133 | 161 | 128
  Grade 3 Headache - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Grade 3 Headache - Dose 1 | 9 | 10 | 10
  Related Headache - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Related Headache - Dose 1 | 104 | 136 | 104
  Any Headache - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Any Headache - Dose 2 | 128 | 129 | 130
  Grade 3 Headache - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Grade 3 Headache - Dose 2 | 14 | 5 | 6
  Related Headache - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Related Headache - Dose 2 | 107 | 108 | 100
  Any Headache - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Any Headache - Dose 3 |  | 124 |
  Grade 3 Headache - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Grade 3 Headache - Dose 3 |  | 11 |
  Related Headache - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Related Headache - Dose 3 |  | 106 |
  Any Headache - Across doses | 204 | 246 | 185
  Grade 3 Headache - Across doses | 19 | 26 | 16
  Related Headache - Across doses | 176 | 219 | 148
  Any Myalgia - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Any Myalgia - Dose 1 | 206 | 236 | 160
  Grade 3 Myalgia - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Grade 3 Myalgia - Dose 1 | 16 | 12 | 8
  Related Myalgia - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Related Myalgia - Dose 1 | 191 | 223 | 140
  Any Myalgia - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Any Myalgia - Dose 2 | 196 | 182 | 150
  Grade 3 Myalgia - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Grade 3 Myalgia - Dose 2 | 13 | 11 | 10
  Related Myalgia - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Related Myalgia - Dose 2 | 182 | 171 | 136
  Any Myalgia - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Any Myalgia - Dose 3 |  | 158 |
  Grade 3 Myalgia - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Grade 3 Myalgia - Dose 3 |  | 8 |
  Related Myalgia - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Related Myalgia - Dose 3 |  | 150 |
  Any Myalgia - Across doses | 278 | 295 | 221
  Grade 3 Myalgia - Across doses | 24 | 25 | 15
  Related Myalgia - Across doses | 265 | 285 | 201
  Any Rash - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Any Rash - Dose 1 | 17 | 8 | 15
  Grade 3 Rash - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Grade 3 Rash - Dose 1 | 1 | 0 | 0
  Related Rash - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Related Rash - Dose 1 | 13 | 5 | 13
  Any Rash - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Any Rash - Dose 2 | 17 | 11 | 16
  Grade 3 Rash - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Grade 3 Rash - Dose 2 | 1 | 0 | 0
  Related Rash - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Related Rash - Dose 2 | 13 | 10 | 16
  Any Rash - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Any Rash - Dose 3 |  | 8 |
  Grade 3 Rash - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Grade 3 Rash - Dose 3 |  | 0 |
  Related Rash - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Related Rash - Dose 3 |  | 5 |
  Any Rash - Across doses | 33 | 25 | 29
  Grade 3 Rash - Across doses | 2 | 0 | 0
  Related Rash - Across doses | 26 | 18 | 28
  Any Fever - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Any Fever - Dose 1 | 24 | 17 | 18
  Grade 3 Fever - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Grade 3 Fever - Dose 1 | 1 | 0 | 0
  Related Fever - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Related Fever - Dose 1 | 15 | 12 | 15
  Any Fever - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Any Fever - Dose 2 | 21 | 15 | 25
  Grade 3 Fever - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Grade 3 Fever - Dose 2 | 1 | 3 | 1
  Related Fever - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Related Fever - Dose 2 | 17 | 12 | 18
  Any Fever - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Any Fever - Dose 3 |  | 29 |
  Grade 3 Fever - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Grade 3 Fever - Dose 3 |  | 0 |
  Related Fever - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Related Fever - Dose 3 |  | 25 |
  Any Fever - Across doses | 41 | 48 | 42
  Grade 3 Fever - Across doses | 2 | 3 | 1
  Related Fever - Across doses | 29 | 39 | 32
  Any Urticaria - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Any Urticaria - Dose 1 | 9 | 7 | 4
  Grade 3 Urticaria - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Grade 3 Urticaria - Dose 1 | 1 | 1 | 0
  Related Urticaria - Dose 1: number analyzed (Participants) | 549 | 480 | 411
  Related Urticaria - Dose 1 | 7 | 3 | 4
  Any Urticaria - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Any Urticaria - Dose 2 | 7 | 9 | 9
  Grade 3 Urticaria - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Grade 3 Urticaria - Dose 2 | 0 | 0 | 0
  Related Urticaria - Dose 2: number analyzed (Participants) | 544 | 470 | 404
  Related Urticaria - Dose 2 | 6 | 7 | 8
  Any Urticaria - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Any Urticaria - Dose 3 |  | 5 |
  Grade 3 Urticaria - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Grade 3 Urticaria - Dose 3 |  | 0 |
  Related Urticaria - Dose 3: number analyzed (Participants) | 0 | 464 | 0
  Related Urticaria - Dose 3 |  | 3 |
  Any Urticaria - Across doses | 15 | 15 | 13
  Grade 3 Urticaria - Across doses | 1 | 1 | 0
  Related Urticaria - Across doses | 13 | 11 | 12

19. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 = unsolicited AE preventing normal activity. Related = unsolicited AE assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 30 day (Days 0-29) post-vaccination period
Population: The analysis was based on the TVC, which included all vaccinated subjects who received at least one dose of vaccine and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group
Number analyzed (Participants) | 550 | 482 | 415
Participants
  Any unsolicited AEs | 97 | 167 | 74
  Grade 3 unsolicited AEs | 2 | 17 | 6
  Related unsolicited AEs | 11 | 24 | 13

20. Secondary Outcome: Number of Subjects With Any Potential Immune-Mediated Diseases (pIMDs)
Description: pIMDs are a subset of AEs that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology.
Time Frame: From Day 0 up to Month 13 (for Cervarix 1 Group and Cervarix 2 Group) and from Day 0 up to Month 18 (for Cervarix 3 Group)
Population: The analysis was based on the TVC, which included all vaccinated subjects who received at least one dose of vaccine and for whom data were available. The data for Cervarix 1 and 2 Groups are only presented up to Month 13, as the data were only collected up to Month 13 for those 2 groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group
Number analyzed (Participants) | 550 | 482 | 415
Participants
  Any pIMDs, from Day 0 up to Month 13 | 2 | 2 | 2
  Any pIMDs, from Day 0 up to Month 18: number analyzed (Participants) | 0 | 0 | 415
  Any pIMDs, from Day 0 up to Month 18 |  |  | 2

21. Secondary Outcome: Number of Subjects With Medically Significant Conditions (MSCs)
Description: MSCs include AEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: From Day 0 up to Month 36 (throughout the study period)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group
Number analyzed (Participants) | 550 | 482 | 415
Participants | 134 | 153 | 87

22. Secondary Outcome: Number of Subjects With Any, Related and Fatal Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity or were a congenital anomaly/birth defect in the offspring of a study subject. Any = any SAE regardless of intensity grade or relation to vaccination.
  Related = SAE assessed by the investigator as causally related to the study vaccination.
Time Frame: From Day 0 up to Month 36 (throughout the study period)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group
Number analyzed (Participants) | 550 | 482 | 415
Participants
  Any SAEs | 20 | 28 | 24
  Related SAEs | 0 | 0 | 1
  Fatal SAEs | 0 | 0 | 0

23. Secondary Outcome: Number of Subjects Reporting Pregnancies and Outcomes of Reported Pregnancies
Description: Outcomes of reported pregnancies were: Ectopic pregnancy, Elective termination NO apparent congenital anomaly (ACA), Live Infant NO ACA, Stillbirth NO ACA.
Time Frame: From Day 0 up to Month 36 (throughout the study period)
Population: The analysis was based on the TVC, which included all subjects with the study vaccine administered and who reported any pregnancies and outcomes of reported pregnancies.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group
Number analyzed (Participants) | 1 | 34 | 1
Participants
  Ectopic pregnancy | 0 | 1 | 0
  Elective termination NO ACA | 0 | 2 | 0
  Live Infant NO ACA | 1 | 30 | 1
  Stillbirth NO ACA | 0 | 1 | 0

24. Secondary Outcome: Number of Subjects Completing the Vaccination Course
Description: The number of subjects completing the vaccination course was assessed as the number of subjects with at least one dose received during the study.
Time Frame: From Day 0 up to Month 13
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group
Number analyzed (Participants) | 550 | 482 | 415
Participants | 550 | 482 | 415

ADVERSE EVENTS:
Time Frame: Solicited symptoms were collected during the 7-day period (Days 0-6) after vaccination.Unsolicited AEs were collected during the 30-day period (Days 0-29) after vaccination. SAEs were collected from Day 0 to Month 36.
Description: The occurrence of reported AEs (all/related) was not available and encoded as equal to the number of subjects affected. For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group
All-Cause Mortality (participants affected / at risk) | 0/550 | 0/482 | 0/415
Serious Adverse Events (participants affected / at risk) | 20/550 | 28/482 | 24/415
Other Adverse Events (participants affected / at risk) | 513/550 | 466/482 | 387/415
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix 1 Group (N=550) | Cervarix 2 Group (N=482) | Cervarix 3 Group (N=415)
Dengue fever (Infections and infestations) | 1 (1) | 4 (4) | 3 (3)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Ectopic pregnancy termination (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Salpingitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Salpingo-oophoritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Synovial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 3 (3) | 5 (5)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cervarix 1 Group (N=550) | Cervarix 2 Group (N=482) | Cervarix 3 Group (N=415)
Nasopharyngitis (Infections and infestations) | 22 (22) | 27 (27) | 14 (14)
Pain (General disorders) | 499 (499) | 461/480 (461) | 381/413 (381)
Redness (General disorders) | 247 (247) | 212/480 (212) | 197/413 (197)
Swelling (General disorders) | 225 (225) | 204/480 (204) | 171/413 (171)
Arthralgia (General disorders) | 111 (111) | 107/480 (107) | 93/413 (93)
Fatigue (General disorders) | 247 (247) | 310/480 (310) | 215/413 (215)
Gastrointestinal symptoms (General disorders) | 98 (98) | 134/480 (134) | 77/413 (77)
Headache (General disorders) | 204 (204) | 246/480 (246) | 185/413 (185)
Myalgia (General disorders) | 278 (278) | 295/480 (295) | 221/413 (221)
Rash (General disorders) | 33 (33) | 25/480 (25) | 29/413 (29)
Fever (General disorders) | 41 (41) | 48/480 (48) | 42/413 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.